CLINICAL TRIAL: NCT01626079
Title: A Clinical Evaluation of the Safety and Effectiveness of the MitraClip® System for the Treatment of Functional Mitral Regurgitation in Symptomatic Heart Failure Subjects (COAPT Recruitment Closed). COAPT CAS (Recruitment Closed)
Brief Title: Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients With Functional Mitral Regurgitation (The COAPT Trial) and COAPT CAS
Acronym: COAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-512
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Mitral Regurgitation; Mitral Valve Regurgitation; Treatment of Functional Mitral Regurgitation in Symptomatic Heart Failure Subjects; Heart Failure
Keywords: Functional Mitral Regurgitation; Mitral Valve Regurgitation; Symptomatic Heart Failure; Functional MR; MitraClip; Mitral Valve Insufficiency; Cardiopulmonary exercise testing; COAPT CAS; COAPT Continued Access Study; MitraClip NT
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Masking Description: 614 in the Randomized Group for COAPT Trial and 162 Subjects in the COAPT CAS Group
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MitraClip System (Experimental): Percutaneous mitral valve repair using MitraClip System
  Interventions: Device: MitraClip System
- Control Group (No Intervention): Patients with mitral regurgitation managed non-surgically based on standard hospital clinical practice.
- COAPT CAS Group (Experimental): Percutaneous mitral valve repair using MitraClip System
  Interventions: Device: MitraClip System

INTERVENTIONS:
Device: MitraClip System — Percutaneous mitral valve repair using MitraClip System
  Other Names: MitraClip device; MitraClip
  Arms: COAPT CAS Group; MitraClip System

SUMMARY:
The purpose of the Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients with Functional Mitral Regurgitation (COAPT) Trial is to confirm the safety and effectiveness of the MitraClip System for the treatment of moderate-to-severe or severe functional mitral regurgitation (FMR) in Symptomatic Heart Failure Subjects who are treated per standard of care and who have been determined by the site's local heart team as not appropriate for mitral valve surgery. This randomized controlled trial will provide the opportunity to strengthen or add labeling claims regarding safety and clinical benefits of the MitraClip System for symptomatic heart failure patients with moderate-to-severe or severe functional mitral regurgitation.

Approximately 610 subjects will be randomized at up to 100 investigational sites with approximately 305 subjects targeted to receive the study device. COAPT study completed recruiting subjects in June 2017.

As part of the COAPT trial, a subset of patients will be registered in the cardiopulmonary exercise (CPX) sub-study. The objective of this sub-study is to evaluate the exercise responses in a sub-cohort of COAPT subjects who receive MitraClip device (Device group) compared to the Control group who do not receive MitraClip device. (Note: the CPX Sub-study subjects will contribute to the analyses of the COAPT primary and secondary endpoints)

As an extension of the COAPT RCT trial, COAPT CAS study will be conducted after COAPT enrollment is complete under the same investigational device exemption (IDE(G120024)). The objective of this study is to evaluate the MitraClip® NT System for the treatment of clinically significant functional mitral regurgitation (FMR) in symptomatic heart failure subjects who are treated per standard of care and who have been determined by the site's local heart team as not appropriate for mitral valve surgery. The anticipated Study Completion Date is July 2024. COAPT CAS completed recruiting subjects in March 2019.

DETAILED DESCRIPTION:
Prospective, randomized, parallel-controlled, multicenter clinical evaluation of the MitraClip device for the treatment of clinically significant functional mitral regurgitation in symptomatic heart failure subjects who are treated per standard of care and who have been determined by the site's local heart team as not appropriate for mitral valve surgery. Eligible subjects will be randomized in a 1:1 ratio to the MitraClip device (Device group) or to no MitraClip device (Control group).

As part of the COAPT trial, a subset of patients (at least 50 up to 100 in total) will be registered in the CPX Sub-study, which is designed as a prospective, randomized (1:1 ratio to the MitraClip or no MitraClip device), parallel-controlled, multicenter study registering approximately 50-100 subjects in up to 50 qualified US sites from the COAPT trial. Subjects registered and randomized in the CPX Sub-study will contribute to the total enrollment approximately of 610 subjects in the COAPT trial. Roll-in subjects will not participate in the CPX Sub-study.

The COAPT CAS study is designed as a prospective, multicenter, single arm, continued access registry study. A maximum of 800 subjects (anticipated) will be registered from up to 75 sites in the United States. The enrollment will end once pre-market approval (PMA) of the proposed expanded indication of MitraClip System is obtained. Active follow-up of patients will be performed through 12 months with scheduled visits at 30 days and 12 months. The national Trans catheter Valve Therapy Registry (TVT Registry) will be used for data collection through 12 months. Annual follow-up data from 2 years through year 5 post-implant will be obtained by linkage to the Centers for Medicare and Medicaid Services (CMS) Claims database.

COAPT CAS data may be used to support the PMA application of the labeling claims for the treatment of moderate to severe or severe FMR in symptomatic heart failure subjects. This single arm registry will provide valuable new information regarding use of the MitraClip® NT System under more "real world" conditions.

COAPT study completed recruiting subjects in June 2017. COAPT CAS completed recruiting subjects in March 2019. A total of 162 subjects were enrolled in the COAPT CAS Group.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic functional MR (≥3+) due to cardiomyopathy of either ischemic or non-ischemic etiology determined by assessment of a qualifying transthoracic echocardiogram (TTE) obtained within 90 days and transesophageal echocardiogram (TEE) obtained within 180 days prior to subject registration, with MR severity based principally on the TTE study, confirmed by the Echocardiography Core Lab (ECL). The ECL may request a transesophageal echocardiogram (TEE) to confirm MR etiology.

   Note: Functional MR requires the presence of global or regional left ventricular wall motion abnormalities, which are believed to be the primary cause of the MR. If a flail leaflet or other evidence of degenerative MR is present, the subject is not eligible even if global or regional left ventricular systolic dysfunction is present.

   Note: Qualifying TTE must be obtained after the subject has been stabilized on optimal therapy including Guideline Directed Medical Therapy (GDMT) and at least 30 days after:
   1. a greater than 100% increase or greater than 50% decrease in dose of GDMT
   2. revascularization and/or implant of Cardiac Resynchronization Therapy device (CRT or CRT-D) or reprogramming of an implanted CRT or CRT-D that results in increased biventricular pacing (from <92% to ≥92%)
2. In the judgment of the HF specialist investigator at the site, the subject has been adequately treated per applicable standards, including for coronary artery disease, left ventricular dysfunction, mitral regurgitation and heart failure (e.g., with cardiac resynchronization therapy, revascularization, and/or GDMT). The Eligibility Committee must also concur that the subject has been adequately treated.
3. New York Heart Association (NYHA) Functional Class II, III or ambulatory IV.
4. The Local Site Heart Team (CT surgeon and HF specialist investigators) and the Central Eligibility Committee concur that surgery will not be offered as a treatment option and that medical therapy is the intended therapy for the subject, even if the subject is randomized to the Control group.
5. The subject has had at least one hospitalization for heart failure in the 12 months prior to subject registration and/or a corrected brain natriuretic peptide (BNP) ≥300 pg/ml or corrected n-Terminal pro- brain natriuretic peptide NT-proBNP ≥1500 pg/ml measured within 90 days prior to subject registration ("corrected" refers to a 4% reduction in the BNP or NT-proBNP cutoff for every increase of 1 kg/m2 in BMI above a reference BMI of 20 kg/m2).

   Note: BNP or NT-proBNP must be obtained after the subject has been stabilized on GDMT and at least 30 days after:
   1. a greater than 100% increase or greater than 50% decrease in dose of GDMT
   2. revascularization and/or implant of Cardiac Resynchronization Therapy device (CRT or CRT-D) or reprogramming of an implanted CRT or CRT-D that results in increased biventricular pacing (from <92% to ≥92%).
6. Left Ventricular Ejection Fraction (LVEF) is ≥20% and ≤50% within 90 days prior to subject registration, assessed by the site using any one of the following methods: echocardiography, contrast left ventriculography, gated blood pool scan or cardiac magnetic resonance imaging (MRI).

   Note: The method must provide a quantitative readout (not a visual assessment).
7. The primary regurgitant jet is non-commissural, and in the opinion of the MitraClip implanting investigator can be successfully be treated by the MitraClip. If a secondary jet exists, it must be considered clinically insignificant.
8. Creatine Kinase-MB (CK-MB) obtained within prior 14 days < local laboratory Upper Limit of Normal (ULN).
9. Transseptal catheterization and femoral vein access is determined to be feasible by the MitraClip implanting investigator.
10. Age 18 years or older.
11. The subject or the subject's legal representative understands and agrees that should he/she be assigned to the Control group, he/she will be treated with medical therapy and conservative management without surgery and without the MitraClip, either domestically or abroad. If the subject would actively contemplate surgery and/or MitraClip if randomized to Control, he/she should not be registered in this trial.
12. The subject or the subject's legal representative has been informed of the nature of the trial and agrees to its provisions, including the possibility of randomization to the Control group and returning for all required post-procedure follow-up visits, and has provided written informed consent.
13. Left Ventricular End Systolic Dimension (LVESD) is ≤ 70 mm assessed by site based on a transthoracic echocardiographic (TTE) obtained within 90 days prior to subject registration.

For the CPX Sub-study: Subjects have to meet the COAPT study eligibility criteria to be registered in the CPX Sub-study.

COAPT CAS study Inclusion Criteria:

1. Subjects must meet all of the above COAPT RCT inclusion criteria, and must have national Medicare coverage by the Centers for Medicare and Medicaid Services (CMS).

Exclusion Criteria:

1. Chronic Obstructive Pulmonary Disease (COPD) requiring continuous home oxygen therapy or chronic outpatient oral steroid use.
2. Untreated clinically significant coronary artery disease requiring revascularization.
3. Coronary artery bypass grafting (CABG) within 30 days prior to subject registration.
4. Percutaneous coronary intervention within 30 days prior to subject registration.
5. Transcatheter aortic valve replacement (TAVR) within 30 days prior to subject registration.
6. Tricuspid valve disease requiring surgery or transcatheter intervention.
7. Aortic valve disease requiring surgery.
8. Cerebrovascular accident within 30 days prior to subject registration.
9. Severe symptomatic carotid stenosis (> 70% by ultrasound).
10. Carotid surgery or stenting within 30 days prior to subject registration.
11. American College of Cardiology /American Heart Association (ACC/AHA) Stage D heart failure.
12. Presence of any of the following:

    * Estimated pulmonary artery systolic pressure (PASP) > 70 mm Hg assessed by site based on echocardiography or right heart catheterization, unless active vasodilator therapy in the cath lab is able to reduce the pulmonary vascular resistance (PVR) to < 3 Wood Units or between 3 and 4.5 Wood Units with v wave less than twice the mean of the pulmonary capillary wedge pressure
    * Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non ischemic etiology
    * Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
    * Hemodynamic instability requiring inotropic support or mechanical heart assistance.
13. Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction as assessed by site.
14. Implant of any Cardiac Resynchronization Therapy (CRT) or Cardiac Resynchronization Therapy with cardioverter-defibrillator (CRT-D) within the last 30days prior to subject registration.
15. Mitral valve orifice area < 4.0 cm2 assessed by site based on a transthoracic echocardiogram (TTE) within 90 days prior to subject registration.
16. Leaflet anatomy which may preclude MitraClip implantation, proper MitraClip positioning on the leaflets or sufficient reduction in MR by the MitraClip. This evaluation is based on transesophageal echocardiogram (TEE) evaluation of the mitral valve within 180 days prior to subject registration and includes:

    * Insufficient mobile leaflet available for grasping with the MitraClip device
    * Evidence of calcification in the grasping area
    * Presence of a significant cleft in the grasping area
    * Lack of both primary and secondary chordal support in the grasping area
    * Leaflet mobility length < 1 cm
17. Hemodynamic instability defined as systolic pressure < 90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
18. Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months.
19. Life expectancy < 12 months due to non-cardiac conditions.
20. Modified Rankin Scale ≥ 4 disability.
21. Status 1 heart transplant or prior orthotopic heart transplantation.
22. Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure.
23. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
24. Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e., noncompliant, perforated).
25. Active infections requiring current antibiotic therapy.
26. Subjects in whom transesophageal echocardiography (TEE) is contraindicated or high risk.
27. Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically.
28. Pregnant or planning pregnancy within next 12 months.

    Note: Female patients of childbearing age should be instructed to use safe contraception (e.g. intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release.
29. Currently participating in an investigational drug or another device study that has not reached its primary endpoint. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
30. Subject belongs to a vulnerable population per investigator's judgment or subject has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures.

For the CPX Sub-study: Subjects who have any contraindications to CPX and are not capable of performing CPX per investigator's assessment should not be registered in the CPX Sub-study.

COAPT CAS study Exclusion Criteria:

1. Subjects must not meet any of the above COAPT RCT exclusion criteria.

.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2024-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mack, MD, Principal Investigator — Baylor Health Care System; Gregg Stone, MD, Principal Investigator — MOUNT SINAI HOSPITAL; William T Abraham, MD, Principal Investigator — The Ohio State University Heart Center; JoAnn Lindenfeld, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (86):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Scottsdale Healthcare Hospitals, Scottsdale, Arizona
  - Scripps Green Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - University California Davis Medical Center, Sacramento, California
  - Kaiser Permanente - San Francisco Hospital, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Mount Sinai Medical Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Hospital Atlanta, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Kansas Hosp Authority, Kansas City, Kansas
  - Via Christi, Wichita, Kansas
  - St. Joseph's Hospital - Lexington, KY, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Foundation for Med Edu And Research, Rochester, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Nebraska Heart Institute Heart Hospital, Lincoln, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - North Shore, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center / New York Presbyterian Hospital, New York, New York
  - NYP Weill Cornell Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of University Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Wormleysburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas Hospital, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Swedish Medical Center Cherry Hill Campus, Seattle, Washington
- Canada (5):
  - St Paul's - Providence Health Care, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - University of Alberta, Edmonton

REFERENCES:
- [Derived] Goel SS, Guha A, Lindenfeld J, Abraham WT, Kar S, Kapadia SR, Little SH, Lim DS, Reardon MJ, Kleiman NS, Aiyer J, Kotinkaduwa LN, Mack MJ, Stone GW. Impact of Natriuretic Peptide and Prior Hospitalization in Patients With Severe Mitral Regurgitation: COAPT Trial. Circ Cardiovasc Interv. 2025 Jul;18(7):e015192. doi: 10.1161/CIRCINTERVENTIONS.125.015192. Epub 2025 May 13. PMID 40357542
- [Derived] Bohra C, Asch FM, Lerakis S, Little SH, Redfors B, Zhou Z, Li Y, Weissman NJ, Grayburn PA, Kar S, Lim DS, Abraham WT, Lindenfeld J, Mack MJ, Bax JJ, Stone GW. Pulmonary Vein Systolic Flow Reversal and Outcomes in Patients From the Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients With Functional Mitral Regurgitation (COAPT) Trial. Struct Heart. 2024 Jun 26;8(5):100333. doi: 10.1016/j.shj.2024.100333. eCollection 2024 Sep. PMID 39290680
- [Derived] Pio SM, Medvedofsky D, Delgado V, Stassen J, Weissman NJ, Grayburn PA, Kar S, Lim DS, Redfors B, Snyder C, Zhou Z, Alu MC, Kapadia SR, Lindenfeld J, Abraham WT, Mack MJ, Asch FM, Stone GW, Bax JJ; COAPT Trial Investigators. Left Atrial Improvement in Patients With Secondary Mitral Regurgitation and Heart Failure: The COAPT Trial. JACC Cardiovasc Imaging. 2024 Sep;17(9):1015-1027. doi: 10.1016/j.jcmg.2024.03.016. Epub 2024 May 22. PMID 38795108
- [Derived] Shahim B, Cohen DJ, Asch FM, Bax J, George I, Ruck A, Ben-Yehuda O, Kar S, Lim DS, Saxon JT, Zhou Z, Lindenfeld J, Abraham WT, Mack MJ, Stone GW. Repeat Mitral Valve Interventions After Transcatheter Edge-to-Edge Repair: The COAPT Trial. Am J Cardiol. 2024 Jul 15;223:7-14. doi: 10.1016/j.amjcard.2024.05.025. Epub 2024 May 23. PMID 38788821
- [Derived] Coisne A, Scotti A, Granada JF, Grayburn PA, Mack MJ, Cohen DJ, Kar S, Lim DS, Lindenfeld J, Bax J, Kotinkaduwa LN, Redfors B, Weissman NJ, Asch FM, Stone GW. Regurgitant volume to LA volume ratio in patients with secondary MR: the COAPT trial. Eur Heart J Cardiovasc Imaging. 2024 Apr 30;25(5):616-625. doi: 10.1093/ehjci/jead328. PMID 38060997
- [Derived] Pio SM, Medvedofsky D, Stassen J, Delgado V, Namazi F, Weissman NJ, Grayburn P, Kar S, Lim DS, Zhou Z, Alu MC, Redfors B, Kapadia S, Lindenfeld J, Abraham WT, Mack MJ, Asch FM, Stone GW, Bax JJ. Changes in Left Ventricular Global Longitudinal Strain in Patients With Heart Failure and Secondary Mitral Regurgitation: The COAPT Trial. J Am Heart Assoc. 2023 Sep 5;12(17):e029956. doi: 10.1161/JAHA.122.029956. Epub 2023 Aug 30. PMID 37646214
- [Derived] Kong J, Zaroff JG, Ambrosy AP, Fitzpatrick JK, Ku IA, Mishell JM, Kotinkaduwa LN, Redfors B, Beohar N, Ailawadi G, Lindenfeld J, Abraham WT, Mack MJ, Kar S, Lim DS, Whisenant BK, Stone GW. Incidence, Predictors, and Outcomes Associated With Worsening Renal Function in Patients With Heart Failure and Secondary Mitral Regurgitation: The COAPT Trial. J Am Heart Assoc. 2023 Jul 18;12(14):e029504. doi: 10.1161/JAHA.123.029504. Epub 2023 Jul 8. PMID 37421291
- [Derived] Vincent F, Redfors B, Kotinkaduwa LN, Kar S, Lim DS, Mishell JM, Whisenant BK, Lindenfeld J, Abraham WT, Mack MJ, Stone GW. Cerebrovascular Events After Transcatheter Edge-to-Edge Repair and Guideline-Directed Medical Therapy in the COAPT Trial. JACC Cardiovasc Interv. 2023 Jun 26;16(12):1448-1459. doi: 10.1016/j.jcin.2023.03.023. PMID 37380226
- [Derived] Scotti A, Coisne A, Granada JF, Driggin E, Madhavan MV, Zhou Z, Redfors B, Kar S, Lim DS, Cohen DJ, Lindenfeld J, Abraham WT, Mack MJ, Asch FM, Stone GW. Impact of Malnutrition in Patients With Heart Failure and Secondary Mitral Regurgitation: The COAPT Trial. J Am Coll Cardiol. 2023 Jul 11;82(2):128-138. doi: 10.1016/j.jacc.2023.04.047. Epub 2023 Jun 9. PMID 37306651
- [Derived] Lindman BR, Asch FM, Grayburn PA, Mack MJ, Bax JJ, Gonzales H, Goel K, Barker CM, Zalawadiya SK, Zhou Z, Alu MC, Weissman NJ, Abraham WT, Lindenfeld J, Stone GW. Ventricular Remodeling and Outcomes After Mitral Transcatheter Edge-to-Edge Repair in Heart Failure: The COAPT Trial. JACC Cardiovasc Interv. 2023 May 22;16(10):1160-1172. doi: 10.1016/j.jcin.2023.02.031. PMID 37225286
- [Derived] Ludwig S, Conradi L, Cohen DJ, Coisne A, Scotti A, Abraham WT, Ben Ali W, Zhou Z, Li Y, Kar S, Duncan A, Lim DS, Adamo M, Redfors B, Muller DWM, Webb JG, Petronio AS, Ruge H, Nickenig G, Sondergaard L, Adam M, Regazzoli D, Garatti A, Schmidt T, Andreas M, Dahle G, Walther T, Kempfert J, Tang GHL, Redwood S, Taramasso M, Praz F, Fam N, Dumonteil N, Obadia JF, von Bardeleben RS, Rudolph TK, Reardon MJ, Metra M, Denti P, Mack MJ, Hausleiter J, Asch FM, Latib A, Lindenfeld J, Modine T, Stone GW, Granada JF; CHOICE-MI and the COAPT Trial Investigators. Transcatheter Mitral Valve Replacement Versus Medical Therapy for Secondary Mitral Regurgitation: A Propensity Score-Matched Comparison. Circ Cardiovasc Interv. 2023 Jun;16(6):e013045. doi: 10.1161/CIRCINTERVENTIONS.123.013045. Epub 2023 May 16. PMID 37194288
- [Derived] Cox ZL, Zalawadiya SK, Simonato M, Redfors B, Zhou Z, Kotinkaduwa L, Zile MR, Udelson JE, Lim DS, Grayburn PA, Mack MJ, Abraham WT, Stone GW, Lindenfeld J. Guideline-Directed Medical Therapy Tolerability in Patients With Heart Failure and Mitral Regurgitation: The COAPT Trial. JACC Heart Fail. 2023 Jul;11(7):791-805. doi: 10.1016/j.jchf.2023.03.009. Epub 2023 Apr 26. PMID 37115135
- [Derived] Stone GW, Abraham WT, Lindenfeld J, Kar S, Grayburn PA, Lim DS, Mishell JM, Whisenant B, Rinaldi M, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Marx SO, Cohen DJ, Asch FM, Mack MJ; COAPT Investigators. Five-Year Follow-up after Transcatheter Repair of Secondary Mitral Regurgitation. N Engl J Med. 2023 Jun 1;388(22):2037-2048. doi: 10.1056/NEJMoa2300213. Epub 2023 Mar 5. PMID 36876756
- [Derived] Shahim B, Cohen DJ, Ben-Yehuda O, Redfors B, Kar S, Lim DS, Arnold SV, Li Y, Lindenfeld J, Abraham WT, Mack MJ, Stone GW. Impact of Peripheral Artery Disease in Patients With Heart Failure Undergoing Transcatheter Mitral Valve Repair: The COAPT Trial. J Am Heart Assoc. 2023 Feb 21;12(4):e028444. doi: 10.1161/JAHA.122.028444. Epub 2023 Feb 8. PMID 36752227
- [Derived] Giustino G, Camaj A, Kapadia SR, Kar S, Abraham WT, Lindenfeld J, Lim DS, Grayburn PA, Cohen DJ, Redfors B, Zhou Z, Pocock SJ, Asch FM, Mack MJ, Stone GW. Hospitalizations and Mortality in Patients With Secondary Mitral Regurgitation and Heart Failure: The COAPT Trial. J Am Coll Cardiol. 2022 Nov 15;80(20):1857-1868. doi: 10.1016/j.jacc.2022.08.803. PMID 36357085
- [Derived] Brener MI, Grayburn P, Lindenfeld J, Burkhoff D, Liu M, Zhou Z, Alu MC, Medvedofsky DA, Asch FM, Weissman NJ, Bax J, Abraham W, Mack MJ, Stone GW, Hahn RT. Right Ventricular-Pulmonary Arterial Coupling in Patients With HF Secondary MR: Analysis From the COAPT Trial. JACC Cardiovasc Interv. 2021 Oct 25;14(20):2231-2242. doi: 10.1016/j.jcin.2021.07.047. PMID 34674862
- [Derived] Kosmidou I, Lindenfeld J, Abraham WT, Rinaldi MJ, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Gaba P, Rogers JH, Shahim B, Redfors B, Zhang Z, Mack MJ, Stone GW. Sex-Specific Outcomes of Transcatheter Mitral-Valve Repair and Medical Therapy for Mitral Regurgitation in Heart Failure. JACC Heart Fail. 2021 Sep;9(9):674-683. doi: 10.1016/j.jchf.2021.04.011. Epub 2021 Aug 11. PMID 34391744
- [Derived] Arnold SV, Stone GW, Jain SS, Mack MJ, Saxon JT, Zhang Z, Lindenfeld J, Abraham WT, Cohen DJ; COAPT Investigators. Prognostic Importance of Health Status Versus Functional Status in Heart Failure and Secondary Mitral Regurgitation. JACC Heart Fail. 2021 Sep;9(9):684-692. doi: 10.1016/j.jchf.2021.04.012. Epub 2021 Aug 11. PMID 34391740
- [Derived] Shahim B, Ben-Yehuda O, Chen S, Redfors B, Madhavan MV, Kar S, Lim DS, Asch FM, Weissman NJ, Cohen DJ, Arnold SV, Liu M, Lindenfeld J, Abraham WT, Mack MJ, Stone GW. Impact of Diabetes on Outcomes After Transcatheter Mitral Valve Repair in Heart Failure: COAPT Trial. JACC Heart Fail. 2021 Aug;9(8):559-567. doi: 10.1016/j.jchf.2021.03.011. PMID 34325886
- [Derived] Kar S, Mack MJ, Lindenfeld J, Abraham WT, Asch FM, Weissman NJ, Enriquez-Sarano M, Lim DS, Mishell JM, Whisenant BK, Rogers JH, Arnold SV, Cohen DJ, Grayburn PA, Stone GW. Relationship Between Residual Mitral Regurgitation and Clinical and Quality-of-Life Outcomes After Transcatheter and Medical Treatments in Heart Failure: COAPT Trial. Circulation. 2021 Aug 10;144(6):426-437. doi: 10.1161/CIRCULATIONAHA.120.053061. Epub 2021 May 27. PMID 34039025
- [Derived] Gertz ZM, Herrmann HC, Lim DS, Kar S, Kapadia SR, Reed GW, Puri R, Krishnaswamy A, Gersh BJ, Weissman NJ, Asch FM, Grayburn PA, Kosmidou I, Redfors B, Zhang Z, Abraham WT, Lindenfeld J, Stone GW, Mack MJ. Implications of Atrial Fibrillation on the Mechanisms of Mitral Regurgitation and Response to MitraClip in the COAPT Trial. Circ Cardiovasc Interv. 2021 Apr;14(4):e010300. doi: 10.1161/CIRCINTERVENTIONS.120.010300. Epub 2021 Mar 15. PMID 33719505
- [Derived] Mack MJ, Lindenfeld J, Abraham WT, Kar S, Lim DS, Mishell JM, Whisenant BK, Grayburn PA, Rinaldi MJ, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Rogers JH, Marx SO, Cohen DJ, Weissman NJ, Stone GW; COAPT Investigators. 3-Year Outcomes of Transcatheter Mitral Valve Repair in Patients With Heart Failure. J Am Coll Cardiol. 2021 Mar 2;77(8):1029-1040. doi: 10.1016/j.jacc.2020.12.047. PMID 33632476
- [Derived] Lindenfeld J, Abraham WT, Grayburn PA, Kar S, Asch FM, Lim DS, Nie H, Singhal P, Sundareswaran KS, Weissman NJ, Mack MJ, Stone GW; Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients With Functional Mitral Regurgitation (COAPT) Investigators. Association of Effective Regurgitation Orifice Area to Left Ventricular End-Diastolic Volume Ratio With Transcatheter Mitral Valve Repair Outcomes: A Secondary Analysis of the COAPT Trial. JAMA Cardiol. 2021 Apr 1;6(4):427-436. doi: 10.1001/jamacardio.2020.7200. PMID 33533873
- [Derived] Saxon JT, Cohen DJ, Chhatriwalla AK, Kotinkaduwa LN, Kar S, Lim DS, Abraham WT, Lindenfeld J, Mack MJ, Arnold SV, Stone GW. Impact of COPD on Outcomes After MitraClip for Secondary Mitral Regurgitation: The COAPT Trial. JACC Cardiovasc Interv. 2020 Dec 14;13(23):2795-2803. doi: 10.1016/j.jcin.2020.09.023. PMID 33303119
- [Derived] Kosmidou I, Lindenfeld J, Abraham WT, Kar S, Lim DS, Mishell JM, Whisenant BK, Kipperman RM, Boudoulas KD, Redfors B, Shahim B, Zhang Z, Mack MJ, Stone GW. Transcatheter Mitral Valve Repair in Patients With and Without Cardiac Resynchronization Therapy: The COAPT Trial. Circ Heart Fail. 2020 Nov;13(11):e007293. doi: 10.1161/CIRCHEARTFAILURE.120.007293. Epub 2020 Nov 12. PMID 33176460
- [Derived] Giustino G, Lindenfeld J, Abraham WT, Kar S, Lim DS, Grayburn PA, Kapadia SR, Cohen DJ, Kotinkaduwa LN, Weissman NJ, Mack MJ, Stone GW. NYHA Functional Classification and Outcomes After Transcatheter Mitral Valve Repair in Heart Failure: The COAPT Trial. JACC Cardiovasc Interv. 2020 Oct 26;13(20):2317-2328. doi: 10.1016/j.jcin.2020.06.058. PMID 33092705
- [Derived] Hahn RT, Asch F, Weissman NJ, Grayburn P, Kar S, Lim S, Ben-Yehuda O, Shahim B, Chen S, Liu M, Redfors B, Medvedofsky D, Puri R, Kapadia S, Sannino A, Lindenfeld J, Abraham WT, Mack MJ, Stone GW. Impact of Tricuspid Regurgitation on Clinical Outcomes: The COAPT Trial. J Am Coll Cardiol. 2020 Sep 15;76(11):1305-1314. doi: 10.1016/j.jacc.2020.07.035. PMID 32912445
- [Derived] Grayburn PA, Sannino A, Cohen DJ, Kar S, Lim DS, Mishell JM, Whisenant BK, Rinaldi MJ, Kapadia SR, Rajagopal V, Crowley A, Kotinkaduwa LN, Lindenfeld J, Abraham WT, Mack MJ, Stone GW. Predictors of Clinical Response to Transcatheter Reduction of Secondary Mitral Regurgitation: The COAPT Trial. J Am Coll Cardiol. 2020 Sep 1;76(9):1007-1014. doi: 10.1016/j.jacc.2020.07.010. PMID 32854834
- [Derived] Arnold SV, Stone GW, Mack MJ, Chhatriwalla AK, Austin BA, Zhang Z, Ben-Yehuda O, Kar S, Lim DS, Lindenfeld J, Abraham WT, Cohen DJ; COAPT Investigators. Health Status Changes and Outcomes in Patients With Heart Failure and Mitral Regurgitation: COAPT Trial. J Am Coll Cardiol. 2020 May 5;75(17):2099-2106. doi: 10.1016/j.jacc.2020.03.002. Epub 2020 Mar 16. PMID 32194195
- [Derived] Tang GHL. Echocardiographic Understanding of Secondary Mitral Regurgitation in Transcatheter Mitral Valve Repair: More to Learn. J Am Coll Cardiol. 2019 Dec 17;74(24):2980-2981. doi: 10.1016/j.jacc.2019.11.001. Epub 2019 Dec 9. No abstract available. PMID 31865965
- [Derived] Asch FM, Grayburn PA, Siegel RJ, Kar S, Lim DS, Zaroff JG, Mishell JM, Whisenant B, Mack MJ, Lindenfeld J, Abraham WT, Stone GW, Weissman NJ; COAPT Investigators. Echocardiographic Outcomes After Transcatheter Leaflet Approximation in Patients With Secondary Mitral Regurgitation: The COAPT Trial. J Am Coll Cardiol. 2019 Dec 17;74(24):2969-2979. doi: 10.1016/j.jacc.2019.09.017. Epub 2019 Sep 28. PMID 31574303
- [Derived] Baron SJ, Wang K, Arnold SV, Magnuson EA, Whisenant B, Brieke A, Rinaldi M, Asgar AW, Lindenfeld J, Abraham WT, Mack MJ, Stone GW, Cohen DJ; COAPT Investigators. Cost-Effectiveness of Transcatheter Mitral Valve Repair Versus Medical Therapy in Patients With Heart Failure and Secondary Mitral Regurgitation: Results From the COAPT Trial. Circulation. 2019 Dec 3;140(23):1881-1891. doi: 10.1161/CIRCULATIONAHA.119.043275. Epub 2019 Sep 29. PMID 31564137
- [Derived] Arnold SV, Chinnakondepalli KM, Spertus JA, Magnuson EA, Baron SJ, Kar S, Lim DS, Mishell JM, Abraham WT, Lindenfeld JA, Mack MJ, Stone GW, Cohen DJ; COAPT Investigators. Health Status After Transcatheter Mitral-Valve Repair in Heart Failure and Secondary Mitral Regurgitation: COAPT Trial. J Am Coll Cardiol. 2019 May 7;73(17):2123-2132. doi: 10.1016/j.jacc.2019.02.010. Epub 2019 Mar 17. PMID 30894288
- [Derived] Stone GW, Lindenfeld J, Abraham WT, Kar S, Lim DS, Mishell JM, Whisenant B, Grayburn PA, Rinaldi M, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Marx SO, Cohen DJ, Weissman NJ, Mack MJ; COAPT Investigators. Transcatheter Mitral-Valve Repair in Patients with Heart Failure. N Engl J Med. 2018 Dec 13;379(24):2307-2318. doi: 10.1056/NEJMoa1806640. Epub 2018 Sep 23. PMID 30280640
- [Derived] Mack MJ, Abraham WT, Lindenfeld J, Bolling SF, Feldman TE, Grayburn PA, Kapadia SR, McCarthy PM, Lim DS, Udelson JE, Zile MR, Gammie JS, Gillinov AM, Glower DD, Heimansohn DA, Suri RM, Ellis JT, Shu Y, Kar S, Weissman NJ, Stone GW. Cardiovascular Outcomes Assessment of the MitraClip in Patients with Heart Failure and Secondary Mitral Regurgitation: Design and rationale of the COAPT trial. Am Heart J. 2018 Nov;205:1-11. doi: 10.1016/j.ahj.2018.07.021. Epub 2018 Aug 1. PMID 30134187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In COAPT, 614 subjects were randomized. Enrollment concluded on June 23, 2017. Of the 614 randomized subjects, 302 were in Device group and 312 in the Control group. Subject follow-up is complete in the COAPT IDE study.
  In COAPT CAS Group, 162 new subjects were enrolled. All 162 subjects received MitraClip device. Enrollment concluded in March 2019. Subject follow-up is on-going in the COAPT CAS study.
  Total enrollment = 614 (COAPT = 302 MitraClip + 314 Control) + 162 (COAPT CAS) = 776
Pre-assignment Details: This section includes the results for the primary safety, primary effectiveness, and the 10 secondary endpoints that are the most essential outcomes of the COAPT trial and also the Primary safety, primary effectiveness and other endpoints for the COAPT CAS Group.
Groups:
- COAPT CAS Group: 162 Subjects enrolled in the COAPT Continued access study (CAS) group.
  Subject follow-up until occurred until 12-month visit.
Period: Overall Study
Arm/Group | MitraClip System | Control Group | COAPT CAS Group
Started | 302 | 312 | 162
Completed | 104 | 75 | 110
Not Completed | 198 | 237 | 52
Not completed — Death | 167 | 192 | 39
Not completed — Withdrawal by Subject | 23 | 37 | 5
Not completed — Lost to Follow-up | 7 | 4 | 2
Not completed — Missed Visits | 1 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Of the 614 subjects, 302 from MitraClip system group and 312 from Control group completed the baseline visit.
  162 subjects enrolled in the COAPT CAS group
Groups:
- COAPT CAS Group: subjects who received Percutaneous mitral valve repair using MitraClip System in the COAPT continued access study (CAS) group.
- Total: Total of all reporting groups
Arm/Group | MitraClip System | Control Group | COAPT CAS Group | Total
Number analyzed (Participants) | 302 | 312 | 162 | 776
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (11.8) | 72.8 (10.5) | 74.5 (10.3) | 72.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 120 | 57 | 278
  Male | 201 | 192 | 105 | 498
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race/Ethnicity: Asian | 6 | 12 | 5 | 23
  Race/Ethnicity: Black or African American | 44 | 44 | 28 | 116
  Race/Ethnicity: Hispanic or Latino | 20 | 20 | 0 | 40
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Race/Ethnicity: White or Caucasian | 225 | 232 | 129 | 586
  Race/Ethnicity: Other | 6 | 4 | 0 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 14 | 0 | 26
  United States | 290 | 298 | 162 | 588
Height [Mean (Standard Deviation); unit: Cm] — Population: Data is missing for 1 subject in Device group and 6 subjects in control group
  Cm
    number analyzed (Participants) | 301 | 306 | 162 | 769
    (all) | 170.84 (10.35) | 169.86 (10.75) | 171.11 (10.38) | 170.34 (10.56)
Weight [Mean (Standard Deviation); unit: Kg] — Population: Data is missing for 1 subject in Device group and 5 subjects in Control group.
  Kg
    number analyzed (Participants) | 301 | 307 | 162 | 770
    (all) | 78.79 (17.23) | 78.40 (20.06) | 79.08 (18.76) | 78.59 (18.70)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: Kg/m^2] — Population: Data is missing for 2 subjects for Device and 7 subjects for Control group.
  Kg/m^2
    number analyzed (Participants) | 301 | 305 | 162 | 768
    (all) | 27.04 (5.81) | 27.05 (5.96) | 26.93 (5.63) | 27.05 (5.88)
Serum Creatinine (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] — Population: Data is missing for 2 subjects in Device group and 6 subjects in Control group.
  (mg/dL)
    number analyzed (Participants) | 300 | 306 | 162 | 768
    (all) | 1.77 (1.22) | 1.80 (1.42) | 1.93 (1.54) | 1.79 (1.32)
Creatinine Clearance (mL/min) [Mean (Standard Deviation); unit: mL/min] — Population: Data is missing for 3 subjects in Device group and 10 subjects in Control group.
  mL/min
    number analyzed (Participants) | 299 | 302 | 162 | 763
    (all) | 50.87 (28.48) | 47.76 (24.97) | 0 (0) | 49.31 (26.79)
Creatinine Clearance <= 60mL/min [Count of Participants; unit: Participants] — Population: Data is missing for 3 subjects in Device group and 10 subjects in Control group
  Participants
    number analyzed (Participants) | 299 | 302 | 162 | 763
    (all) | 214 | 227 | 0 | 441
Brain Natriuretic Peptide (Pg/mL) [Mean (Standard Deviation); unit: Pg/mL] — Population: Not all subjects had Brain Natriuretic Peptide (BNP) value collected. some subjects were on NT-proBNP.
  Pg/mL
    number analyzed (Participants) | 208 | 209 | 162 | 579
    (all) | 1014.77 (1085.98) | 1017.13 (1212.77) | 1224.2 (1270.4) | 1015.95 (1149.89)
NT-proBNP (pg/mL) [Mean (Standard Deviation); unit: pg/mL] — Population: Majority of subjects had BNP available. Subjects who did not have BNP had NT-proBNP available.
  pg/mL
    number analyzed (Participants) | 74 | 85 | 162 | 321
    (all) | 5174.33 (6566.61) | 5943.86 (8437.61) | 6885.3 (8287.0) | 5585.71 (7610.56)
Elevated BNP or NT-BNP prior to Enrollment [Count of Participants; unit: Participants] — Population: All available data reported
  Participants
    number analyzed (Participants) | 286 | 303 | 162 | 751
    (all) | 267 | 282 | 0 | 549
Extremely High Risk for MV Surgery [Count of Participants; unit: Participants] — High surgical risk if investigational site assessed a predicted surgical mortality for mitral valve surgery of ≥ 12% based on either:
  I) STS (Society of Thoracic Surgeons) mortality risk ≥ 12%, or
  II) The presence of at least one of the following:
  1. Porcelain aorta or mobile ascending aortic atheroma
  2. Post-radiation mediastinum
  3. Previous mediastinitis
  4. Functional MR with EF < 40%
  5. Over 75 years old with EF < 40%
  6. Prior re-operation with patent grafts
  7. Two or more prior chest surgeries
  8. Hepatic cirrhosis
  9. Three or more of the following STS high risk factors Population: Not all subjects met the criteria for High Risk for MV Surgery
  Participants
    number analyzed (Participants) | 299 | 312 | 162 | 773
    (all) | 205 | 218 | 0 | 423
Diabetes [Count of Participants; unit: Participants] | 106 | 123 | 51 | 280
Hypertension [Count of Participants; unit: Participants] | 243 | 251 | 137 | 631
Hypercholesterolemia [Count of Participants; unit: Participants] | 166 | 163 | 0 | 329
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 156 | 160 | 65 | 381
Previous Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 130 | 153 | 63 | 346
Previous Coronary Artery Bypass Grafting [Count of Participants; unit: Participants] | 121 | 126 | 51 | 298
Previous Stroke or Transient Ischemic Attack [Count of Participants; unit: Participants] | 56 | 49 | 9 | 114
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 52 | 57 | 34 | 143
Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] | 71 | 72 | 0 | 143
History of Atrial Fibrillation or Flutter [Count of Participants; unit: Participants] | 173 | 166 | 99 | 438
Anemia [Count of Participants; unit: Participants] — Population: All available data is reported
  Participants
    number analyzed (Participants) | 301 | 306 | 162 | 769
    (all) | 180 | 192 | 0 | 372
STS Risk Score [Mean (Standard Deviation); unit: percentage of expected mortality] — The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk.
  As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries.
  percentage of expected mortality | 7.83 (5.53) | 8.5 (6.15) | 9.26 (6.39) | 8.17 (5.86)
STS Risk Score >= 8% [Count of Participants; unit: Participants] — The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk.
  As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries.
  Participants | 126 | 136 | 78 | 340
Risk of Surgery-related complications or death [Count of Participants; unit: Participants] — Subjects were evaluated by the Local Site Heart Team based on their medical history to determine their risk of surgery related complications or death. Population: All available data is reported
  Participants
    High: number analyzed (Participants) | 299 | 312 | 162 | 773
    High | 205 | 218 | 0 | 423
    Not High: number analyzed (Participants) | 299 | 312 | 162 | 773
    Not High | 94 | 94 | 0 | 188
Cardiomyopathy [Count of Participants; unit: Participants]
  Ischemic | 184 | 189 | 73 | 446
  Non-Ischemic | 118 | 123 | 66 | 307
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms Class IV - Severe limitations.
  Participants
    NYHA Class I | 1 | 0 | 0 | 1
    NYHA Class II | 129 | 110 | 30 | 269
    NYHA Class III | 154 | 168 | 111 | 433
    NYHA Class IVa, ambulatory | 18 | 33 | 21 | 72
Hospitalization for Heart Failure within Previous 1 yr [Count of Participants; unit: Participants] | 176 | 175 | 105 | 456
Previous Cardiac Resynchronization Therapy [Count of Participants; unit: Participants] | 115 | 109 | 25 | 249
Previous Implantation of Defibrillator [Count of Participants; unit: Participants] | 91 | 101 | 95 | 287
Severity of Mitral Regurgitation [Count of Participants; unit: Participants] — Population: In the Control group, baseline echocardiography data was not readable. Hence 311 participants were analyzed.
  Participants
    Moderate-to-severe, grade 3+: number analyzed (Participants) | 302 | 311 | 162 | 775
    Moderate-to-severe, grade 3+ | 148 | 172 | 54 | 374
    Severe, grade 4+: number analyzed (Participants) | 302 | 311 | 162 | 775
    Severe, grade 4+ | 154 | 139 | 99 | 392
Effective Regurgitat Orifice Area [Mean (Standard Deviation); unit: Cm2] — Population: EROA was not measurable for all subjects
  Cm2
    number analyzed (Participants) | 289 | 302 | 162 | 753
    (all) | 0.41 (0.15) | 0.40 (0.15) | 0.70 (1.16) | 0.41 (0.15)
Left Ventricular End Systolic Dimension (Diameter) [Mean (Standard Deviation); unit: cm] — left ventricle end-systolic diameter, is measured at end systole, on the frame preceding mitral valve opening. It corresponds to the smallest cardiac dimension. Population: LVESD was not measurable for all subjects
  cm
    number analyzed (Participants) | 301 | 306 | 162 | 769
    (all) | 5.28 (0.86) | 5.30 (0.89) | 1.16 (0.95) | 5.29 (0.87)
Left Ventricular End-Diastolic Dimension [Mean (Standard Deviation); unit: cm] — Population: LVEDD was not measurable in all subjects
  cm
    number analyzed (Participants) | 301 | 307 | 162 | 770
    (all) | 6.17 (0.73) | 6.19 (0.75) | 6.23 (0.86) | 6.18 (0.74)
Left Ventricular End-Systolic Volume [Mean (Standard Deviation); unit: mL] — Population: LVESV was not measurable for all subjects
  mL
    number analyzed (Participants) | 281 | 294 | 162 | 737
    (all) | 135.5 (56.1) | 134.3 (60.3) | 132.3 (65.4) | 134.9 (58.2)
Left Ventricular End-Diastolic Volume [Mean (Standard Deviation); unit: mL] — Population: LVEDV was not measurable in all subjects
  mL
    number analyzed (Participants) | 281 | 294 | 162 | 737
    (all) | 194.4 (69.2) | 191.0 (72.9) | 185.8 (81.2) | 192.7 (71.0)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: %] — Population: LVEF was not measured for all subjects
  %
    number analyzed (Participants) | 281 | 294 | 162 | 737
    (all) | 31.32 (9.07) | 31.30 (9.58) | 32.2 (9.9) | 31.31 (9.32)
LVEF >= 40% [Count of Participants; unit: Participants] — Population: All available data is reported
  Participants
    number analyzed (Participants) | 281 | 294 | 162 | 737
    (all) | 231 | 241 | 28 | 500
Right Ventricular Systolic Pressure [Mean (Standard Deviation); unit: mmHg] — Population: All available data is reported
  mmHg
    number analyzed (Participants) | 253 | 275 | 162 | 690
    (all) | 43.95 (13.44) | 44.56 (13.96) | 0 (0) | 44.26 (13.70)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Percentage of Participants With Freedom From Device Related Complications at 12 Months
Description: Percentage of Participants with Freedom from Device related Complications at 12 Months.
  Composite of Single Leaflet Device Attachment (SLDA), device embolizations, endocarditis requiring surgery, Echocardiography Core Laboratory confirmed mitral stenosis requiring surgery, LVAD implant, heart transplant, and any device related complications requiring non-elective cardiovascular surgery.
Time Frame: 12 months
Population: Subjects who were randomized with attempted procedure to the device group with available data. Performance goal was 88%.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 293
percentage of participants | 0.966 [0.948 to NA] — Upper limit is NA as this is a one sided 95% confidence interval.
Statistical Analysis 1: Comparison: MitraClip System; Test type: Non-Inferiority — Two thousand (2000) simulations were performed to calculate sample size and power for the primary safety endpoint. Assuming 22% mortality and 7.5% attrition at 12 months, a total of 305 subjects in the Device group will provide > 95% power to reject the null hypothesis at the one-sided significance level of 5%; p < 0.0001, Z test Using Kaplan Meier Survival; P-value calculated from Z test using Kaplan Meier survival estimate together with Greenwood method estimated variance; Kaplan Meier = 0.966, 95% CI 1-sided [lower limit 0.948], Standard Error of Mean 0.011

2. Primary Outcome: Primary Effectiveness Endpoint
Description: Recurrent HF hospitalizations (HFH) through 24 months, analyzed when the last subject completes 12-month follow-up
Time Frame: 24 months
Population: 302 subjects from device group and 312 subjects from the control group were analyzed for Recurrent HF hospitalizations through 24 months
Measure: Number; unit: events
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
events | 160 | 283

3. Primary Outcome: Primary Effectiveness Endpoint
Description: Recurrent HF hospitalizations (HFH) through 24 months, analyzed when the last subject completes 12-month follow-up
Time Frame: 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 92 | 151

4. Secondary Outcome: Recurrent Heart Failure (HF) Hospitalization (COAPT CAS Study Analysis)
Description: Number of recurrent Heart Failure hospitalization events at 12 months.
Time Frame: 12 months
Population: A total of 162 subjects were enrolled in the COAPT CAS study.
Measure: Number; unit: Events
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Events | 52

5. Secondary Outcome: New York Heart Association (NYHA) Functional Class (COAPT CAS Study Analysis)
Description: The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms Class IV - Severe limitations.
Time Frame: 12 months
Population: A total of 162 subjects were enrolled in the COAPT CAS study. Of them NYHA data was available for a total of 93 subjects at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 93
Participants
  NYHA Class I | 21
  NYHA Class II | 44
  NYHA Class III | 23
  NYHA Class IV | 5

6. Secondary Outcome: New York Heart Association (NYHA) Functional Class (COAPT CAS Study Analysis)
Description: as for outcome 5
Time Frame: 30 days
Population: A total of 162 subjects were enrolled in the COAPT CAS study. Of them NYHA data was available for a total of 142 subjects at 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 142
Participants
  NYHA Class I | 30
  NYHA Class II | 66
  NYHA Class III | 43
  NYHA Class IV | 3

7. Secondary Outcome: Quality of Life (QOL) (COAPT CAS Study Analysis) Quality of Life (QoL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The Kansas City Cardiomyopathy Questionnaire is a 23-item, self administered instrument that quantifies physicalfunction, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possiblesubscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies thefollowing six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical FunctionDomain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQSymptom Stability Domain, Clinical Summary Score and Overall Summary Score. Clinical Summary Scoreincludes total symptom and physical function scores to correspond with NYHA Classification. Overall SummaryScore includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: 12 months
Population: A total of 162 subjects were enrolled in the COAPT CAS study. Data was available for 93 subjects at 12 months.
Measure: Mean (Standard Deviation); unit: KCCQ Score on a points scale
Arm/Group | MitraClip System
Number analyzed (Participants) | 93
KCCQ Score on a points scale | 65.93 (23.80)

8. Secondary Outcome: Quality of Life (QOL) (COAPT CAS Study Analysis) Quality of Life (QoL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The Kansas City Cardiomyopathy Questionnaire is a 23-item, self administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score. Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification. Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: 30 days
Population: A total of 162 subjects were enrolled in the COAPT CAS study. Data was available for 143 subjects at 30 days.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System
Number analyzed (Participants) | 143
KCCQ score on a points scale | 61.36 (25.00)

9. Secondary Outcome: Six Minute Walk Test (6MWT Distance or 6MWD) (COAPT CAS Study Analysis)
Description: The Six Minute Walk Test (6MWT) is a practical simple test that requires a 100-ft hallway but no exerciseequipment or advanced training for technicians. This test measures the distance that a patient can quickly walk ona flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of allthe systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation,peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific informationon the function of each of the different organs and systems involved in exercise or the mechanism of exerciselimitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses thesubmaximal level of functional capacity.
Time Frame: 12 months
Population: A total of 162 subjects were enrolled in the COAPT CAS study. 6MWT data was available for 72 subjects at 12 months.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System
Number analyzed (Participants) | 72
meters | 219.87 (124.82)

10. Secondary Outcome: Six Minute Walk Test (6MWT Distance or 6MWD) (COAPT CAS Study Analysis)
Description: The Six Minute Walk Test (6MWT) is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity.
Time Frame: 30 days
Population: A total of 162 subjects were enrolled in the COAPT CAS study. 6MWT data was available for 117 subjects at 30 days..
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System
Number analyzed (Participants) | 117
meters | 231.24 (145.98)

11. Secondary Outcome: Mitral Regurgitation (MR) Severity (COAPT CAS Study Analysis)
Description: MR Severity Grading was done by Quantitative Doppler Echocardiography and subjects were graded as below MR 1+ - Regurgitant Volume < 30 ml, Right ventricular EF <30%, Effective regurgitant orifice area < 20 mm^2 MR2+ - Regurgitant Volume 30-44 ml, Right ventricular EF 30-39%, Effective regurgitant orifice area 20-29 mm^2 MR3+ - Regurgitant Volume 45-59 ml, Right ventricular EF 40-49 %, Effective regurgitant orifice area 30-39 mm^2MR 4+ - Regurgitant Volume >= 60 ml, Right ventricular EF >=50%, Effective regurgitant orifice area >=40 mm^2
Time Frame: 12 months
Population: Echocardiogram data was available for 98 subjects at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 98
Participants
  None or Trace/Trivial | 9
  Mild (1+) | 53
  Moderate (2+) | 27
  Moderate - Severe (3+) | 6
  Severe (4+) | 3

12. Secondary Outcome: Mitral Regurgitation (MR) Severity (COAPT CAS Study Analysis)
Description: MR Severity Grading was done by Quantitative Doppler Echocardiography and subjects were graded as below
  MR 1+ - Regurgitant Volume < 30 ml, Right ventricular EF <30%, Effective regurgitant orifice area < 20 mm^2 MR 2+ - Regurgitant Volume 30-44 ml, Right ventricular EF 30-39%, Effective regurgitant orifice area 20-29 mm^2 MR 3+ - Regurgitant Volume 45-59 ml, Right ventricular EF 40-49 %, Effective regurgitant orifice area 30-39 mm^2 MR 4+ - Regurgitant Volume >= 60 ml, Right ventricular EF >=50%, Effective regurgitant orifice area >=40 mm^2
Time Frame: 30 days
Population: Echocardiogram data was available for 149 subjects at 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 149
Participants
  None or Trace/Trivial | 11
  Mild (1+) | 85
  Moderate (2+) | 40
  Moderate - Severe (3+) | 9
  Severe (4+) | 4

13. Secondary Outcome: Major and/or Life Threatening Bleeding (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 4

14. Secondary Outcome: Major and/or Life Threatening Bleeding (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 1

15. Secondary Outcome: Major Vascular Complications (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 1

16. Secondary Outcome: Major Vascular Complications (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 0

17. Secondary Outcome: Renal Complication With Requirement for Dialysis (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 4

18. Secondary Outcome: Renal Complication With Requirement for Dialysis (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 2

19. Secondary Outcome: Transient Ischemic Attack (TIA) (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 0

20. Secondary Outcome: Transient Ischemic Attack (TIA) (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 0

21. Secondary Outcome: Stroke (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 1

22. Secondary Outcome: Stroke (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 1

23. Secondary Outcome: Myocardial Infarction (MI) (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 0

24. Secondary Outcome: Myocardial Infarction (MI) (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants | 0

25. Secondary Outcome: Death and Primary Cause of Death (COAPT CAS Study Analysis)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants
  Cardiac | 13
  Neurologic | 2
  Renal | 0
  Vascular | 0
  Infection | 1
  Valvular | 0
  Unknown | 24
  Other | 1
  Not Available | 1

26. Secondary Outcome: Death and Primary Cause of Death (COAPT CAS Study Analysis)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 162
Participants
  Cardiac | 2
  Neurologic | 0
  Renal | 0
  Vascular | 0
  Infection | 0
  Valvular | 0
  Unknown | 1
  Other | 0

27. Secondary Outcome: Percentage of Patients Free From the Composite of All-cause Death, Stroke, MI, or Non-elective Cardiovascular Surgery for Device Related Complications in the Device Group
Description: The percentage of patients free from the composite endpoint as described above.
Time Frame: 30 days post-procedure in the Device group
Population: All device subjects
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 302
Percentage of Participants | 96.9 [94.7 to 96.9]

28. Secondary Outcome: Number of Deaths at 12 Months (All Cause Mortality)
Description: Death from any cause mortality at 12months.
Time Frame: 12 months
Population: All device and control group subjects were included in the analysis.
Measure: Number; unit: participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
participants | 57 | 70

29. Secondary Outcome: Number of Participants With Mitral Regurgitation Severity Grade of 2+ or Lower at 12 Months
Description: MR severity grade of 2+ or lower at 12 months MR Severity Grading was done by Quantitative Doppler Echocardiography and subjects were graded as below
  MR 1+ - Regurgitant Volume < 30 ml, Right ventricular EF <30%, Effective regurgitant orifice area < 20 mm^2 MR 2+ - Regurgitant Volume 30-44 ml, Right ventricular EF 30-39%, Effective regurgitant orifice area 20-29 mm^2 MR 3+ - Regurgitant Volume 45-59 ml, Right ventricular EF 40-49 %, Effective regurgitant orifice area 30-39 mm^2 MR 4+ - Regurgitant Volume >= 60 ml, Right ventricular EF >=50%, Effective regurgitant orifice area >=40 mm^2
Time Frame: 12 months
Population: Echocardiography data was available for 210 subjects in Device group and 175 subjects in Control group
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 210 | 175
Participants | 199 | 82

30. Secondary Outcome: Change in Distance Walked on the 6 Minute Walk Test (6MWT Distance or 6MWD)
Description: The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity.
Time Frame: 12 months over baseline
Population: Analysis population includes subjects still active and with paired available compared to baseline.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 230 | 237
meters | -2.17 (9.12) | -60.2 (8.99)

31. Secondary Outcome: Change in Quality of Life (QoL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Paired data looking at difference between the baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) and 12 month KCCQ score.
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score.
  Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification.
  Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: 12 months over baseline
Population: Analysis population includes subjects still active and with paired available compared to baseline.
Measure: Mean (Standard Deviation); unit: KCCQ Score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 237 | 228
KCCQ Score on a points scale | 12.5 (1.8) | -3.6 (1.9)

32. Secondary Outcome: Change in Left Ventricular End Diastolic Volume (LVEDV)
Description: Paired data comparing the Change in LVEDV at baseline vs 12 months
Time Frame: 12 months over baseline
Population: Analysis population includes subjects with echocardiography paired data available
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 175 | 174
mL | -3.71 (5.08) | 17.06 (5.10)

33. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class I/II
Description: NEW YORK HEART ASSOCIATION CLASSIFICATION (NYHA CLASS)
  Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. Patients are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 12 months
Population: Analysis population includes subjects with available NYHA class data at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 237 | 232
Participants | 171 | 115

34. Secondary Outcome: Recurrent Hospitalizations - All Cause
Description: Number of Recurrent Hospitalizations for any cause within 24 months.
Time Frame: 24 Months
Population: All randomized subjects in Device and Control Group
Measure: Number; unit: Number of Events
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Number of Events | 474 | 610
Statistical Analysis 1: Comparison: MitraClip System vs Control Group; Test type: Superiority; p < 0.02, Joint Fraility Model; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.60 to 0.96]

35. Secondary Outcome: Death or HF Hospitalization Within 24 Months (Finkelstein-Schoenfeld Analysis of All-Cause Death or Recurrent HF Hospitalization Through 24 Months)
Description: The win ratio is a useful method for providing an estimate of the treatment effect when composite endpoints are analyzed as the analysis accounts for clinical significance of the outcomes of interest. For example, in the composite of death and recurrent HF hospitalizations through 24 months, subjects in the Device and Control groups were formed into matched pairs, where each pair of subjects was classified into 1 of 5 outcomes scenarios:
  A. Death in Device group first B. Death in Control group first C. More HF hospitalizations in the Device group (or in the case of a tie, the first HF hospitalization in the Device group occurs first) D. More HF hospitalization in the Control group (or in the case of tie, the first HF hospitalization in the Control group occurs first) E. None of the above In this way, the number of "Winners" in the Device group was NW = NB + ND while the number of "Losers" in the Device group was NL = NA + NC. The "Win Ratio" was then calculated as NW/NL.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Win Ratio
Groups:
- Randomized Group: Randomized group contains both Device and Control Group
Arm/Group | Randomized Group
Number analyzed (Participants) | 614
Win Ratio | 1.61 [1.29 to 2.04]
Statistical Analysis 1: Comparison: Randomized Group; Test type: Superiority; p < 0.0001, Finkelstein-Schoenfeld Analysis; Win Ratio = 1.61, 95% CI 2-sided [1.29 to 2.04]

36. Secondary Outcome: Death and Primary Cause of Death (COAPT CAS Study Analysis)
Description: The COAPT study is still on-going. Only the Primary and major secondary endpoints have been entered. Rest of the results will be entered when the study ends in July 2024.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2024-07

37. Secondary Outcome: Death and Primary Cause of Death (COAPT CAS Study Analysis)
Time Frame: 3 years
Reporting Status: Not Posted

38. Secondary Outcome: Death and Primary Cause of Death (COAPT CAS Study Analysis)
Time Frame: 4 years
Reporting Status: Not Posted

39. Secondary Outcome: Death and Primary Cause of Death (COAPT CAS Study Analysis)
Time Frame: 5 years
Reporting Status: Not Posted

40. Secondary Outcome: Myocardial Infarction (MI) (COAPT CAS Study Analysis)
Time Frame: 2 years
Reporting Status: Not Posted

41. Secondary Outcome: Myocardial Infarction (MI) (COAPT CAS Study Analysis)
Time Frame: 3 years
Reporting Status: Not Posted

42. Secondary Outcome: Myocardial Infarction (MI) (COAPT CAS Study Analysis)
Time Frame: 4 years
Reporting Status: Not Posted

43. Secondary Outcome: Myocardial Infarction (MI) (COAPT CAS Study Analysis)
Time Frame: 5 years
Reporting Status: Not Posted

44. Secondary Outcome: Stroke (COAPT CAS Study Analysis)
Time Frame: 2 years
Reporting Status: Not Posted

45. Secondary Outcome: Stroke (COAPT CAS Study Analysis)
Time Frame: 3 years
Reporting Status: Not Posted

46. Secondary Outcome: Stroke (COAPT CAS Study Analysis)
Time Frame: 4 years
Reporting Status: Not Posted

47. Secondary Outcome: Stroke (COAPT CAS Study Analysis)
Time Frame: 5 years
Reporting Status: Not Posted

48. Secondary Outcome: Recurrent Heart Failure (HF) Hospitalization (COAPT CAS Study Analysis)
Time Frame: 2 years
Reporting Status: Not Posted

49. Secondary Outcome: Recurrent Heart Failure (HF) Hospitalization (COAPT CAS Study Analysis)
Time Frame: 3 years
Reporting Status: Not Posted

50. Secondary Outcome: Recurrent Heart Failure (HF) Hospitalization (COAPT CAS Study Analysis)
Time Frame: 4 years
Reporting Status: Not Posted

51. Secondary Outcome: Recurrent Heart Failure (HF) Hospitalization (COAPT CAS Study Analysis)
Time Frame: 5 years
Reporting Status: Not Posted

52. Secondary Outcome: Kaplan-Meier Freedom From All-cause Mortality
Description: Death from any cause within 24 months - no of events
Time Frame: 24 months
Population: Total number of subjects randomized in the Device and Control group
Measure: Number; unit: no of events
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
no of events | 83 | 125

53. Other Pre Specified Outcome: Device or Procedure-Related Adverse Events
Description: Device or procedure-related adverse events are defined as adverse events that are adjudicated by the Clinical Events Committee as possibly, probably or definitely device and/or procedure-related, regardless of the temporal relationship to the MitraClip procedure. Device or procedure-related adverse events will be broken down into those that occur within 30 days of the procedure and those that occur after 30 days of the procedure. Examples of device-related adverse events are: myocardial perforation, Single Leaflet Device Attachment, embolization of the MitraClip device or MitraClip System components, iatrogenic atrial septal defect, mitral valve stenosis, need for mitral valve replacement instead of repair due at least in part to the MitraClip procedure or the presence of the MitraClip device.
Time Frame: Within and after 30 days of the procedure
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 302
Participants
  Occurred within 30 days | 17
  Occurred between 31 days and 365 days | 4

54. Other Pre Specified Outcome: Implant Rate
Description: Defined as the rate of successful delivery and deployment of the MitraClip device(s) with echocardiographic evidence of leaflet approximation and retrieval of the delivery catheter
Time Frame: Day 0
Population: Subjects randomized to the device arm
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System
Number analyzed (Participants) | 302
Participants | 287

55. Other Pre Specified Outcome: Device Procedure Time
Description: Defined as the time elapsed from the start of the transseptal procedure to the time the Steerable Guide Catheter is removed
Time Frame: Day 0
Population: Device procedure time was not available for all implanted subjects. Data was available for 282 subjects from 302 randomized subjects in device arm.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MitraClip System
Number analyzed (Participants) | 282
minutes | 118.9 (63.5)

56. Other Pre Specified Outcome: Total Procedure Time
Description: Defined as the time elapsed from the first of any of the following: intravascular catheter placement, anesthesia or sedation, or transesophageal echocardiogram (TEE), to the removal of the last catheter and TEE
Time Frame: Day 0
Population: Total procedure time was available for 293 subjects from the 302 subjects randomized to device arm.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MitraClip System
Number analyzed (Participants) | 293
minutes | 162.9 (118.1)

57. Other Pre Specified Outcome: Device Time
Description: Defined as the time the Steerable Guide Catheter is placed in the intra-atrial septum until the time the MitraClip Delivery System (CDS) is retracted into the Steerable Guide Catheter
Time Frame: Day 0
Population: Device time available for all 287 subjects implanted with MitraClip.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MitraClip System
Number analyzed (Participants) | 287
minutes | 82.7 (80.8)

58. Other Pre Specified Outcome: Fluoroscopy Duration
Description: Defined as the duration of exposure to fluoroscopy during the MitraClip procedure
Time Frame: Day 0
Population: Fluoroscopy duration for all available subjects with MitraClip device
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MitraClip System
Number analyzed (Participants) | 284
minutes | 33.9 (23.2)

59. Other Pre Specified Outcome: MR Severity Grade
Description: as for outcome 12
Time Frame: Baseline
Population: echocardiogram data was available for 302 subjects in the device arm and 311 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 311
Participants
  MR 3+ | 148 | 172
  MR 4+ | 154 | 139

60. Other Pre Specified Outcome: MR Severity Grade
Description: as for outcome 12
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: Echocardiogram data was available for 286 subjects in the device arm and 257 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 286 | 257
Participants
  MR None or 1+ | 230 | 21
  MR 2+ | 39 | 67
  MR 3+ | 13 | 96
  MR 4+ | 4 | 73

61. Other Pre Specified Outcome: MR Severity Grade
Description: as for outcome 12
Time Frame: 6 months
Population: Echocardiogram data was available for only 240 subjects in the device group and 218 subjects in the control group
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 240 | 218
Participants
  MR none or 1+ | 160 | 20
  MR 2+ | 65 | 63
  MR 3+ | 11 | 92
  MR 4+ | 4 | 43

62. Other Pre Specified Outcome: MR Severity Grade
Description: as for outcome 12
Time Frame: 12 months
Population: Echocardiogram data was available for 210 subjects in the device arm and 175 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 210 | 175
Participants
  MR None or 1+ | 145 | 20
  MR 2+ | 54 | 62
  MR 3+ | 9 | 60
  MR 4+ | 2 | 33

63. Other Pre Specified Outcome: MR Severity Grade
Description: as for outcome 12
Time Frame: 24 months
Population: Echocardiogram data was available for 167 subjects in the device arm and 126 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 167 | 126
Participants
  MR None or 1+ | 131 | 23
  MR 2+ | 35 | 36
  MR 3+ | 0 | 43
  MR 4+ | 1 | 24

64. Other Pre Specified Outcome: MR Severity Grade
Description: as for outcome 11
Time Frame: 3 years
Population: Echocardiogram data was available for 120 subjects in the device arm and 74 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 120 | 74
Participants
  MR None or 1+ | 100 | 48
  MR 2+ | 18 | 15
  MR 3+ | 2 | 8
  MR 4+ | 0 | 3

65. Other Pre Specified Outcome: MR Severity Grade
Description: MR Severity Grading was done by Quantitative Doppler Echocardiography and subjects were graded as below MR 1+ - Regurgitant Volume < 30 ml, Right ventricular EF <30%, Effective regurgitant orifice area < 20 mm^2 MR 2+ - Regurgitant Volume 30-44 ml, Right ventricular EF 30-39%, Effective regurgitant orifice area 20-29 mm^2 MR 3+ -Regurgitant Volume 45-59 ml, Right ventricular EF 40-49 %, Effective regurgitant orifice area 30-39 mm^2 MR 4+ - Regurgitant Volume >= 60 ml, Right ventricular EF >=50%, Effective regurgitant orifice area >=40 mm^2
Time Frame: 4 years
Population: Echocardiogram data was available for 80 subjects in the device arm and 49 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Groups:
- Device Group: MitraClip Device
- Control Group: Control group treated with medication
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 80 | 49
Participants
  MR None or 1+ | 64 | 30
  MR 2+ | 14 | 9
  MR 3+ | 2 | 6
  MR 4+ | 0 | 4

66. Other Pre Specified Outcome: MR Severity Grade
Description: MR Severity Grading was done by Quantitative Doppler Echocardiography andsubjects were graded as below MR 1+ - Regurgitant Volume < 30 ml, Right ventricular EF <30%, Effectiveregurgitant orifice area < 20 mm^2 MR 2+ - Regurgitant Volume 30-44 ml, Rightventricular EF 30-39%, Effective regurgitant orifice area 20-29 mm^2 MR 3+ -Regurgitant Volume 45-59 ml, Right ventricular EF 40-49 %, Effective regurgitantorifice area 30-39 mm^2 MR 4+ - Regurgitant Volume >= 60 ml, Right ventricularEF >=50%, Effective regurgitant orifice area >=40 mm^2
Time Frame: 5 years
Population: Echocardiogram data was available for 57 subjects in the device arm and 46 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 57 | 46
Participants
  MR None or 1+ | 51 | 36
  MR 2+ | 3 | 6
  MR 3+ | 3 | 2
  MR 4+ | 0 | 2

67. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: Baseline
Population: Echocardiogram data was available for the 289 subjects in the device arm and 302 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 289 | 302
cm^2 | 0.41 (0.15) | 0.40 (0.15)

68. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: Echocardiogram data was available for 75 subjects in the device arm and 73 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 75 | 73
cm^2 | 0.14 (0.08) | 0.23 (0.16)

69. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: 6 months
Population: Echocardiogram data was available for 39 subjects in the device arm and 54 subjects in the control arm
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 39 | 54
cm^2 | 0.22 (0.19) | 0.25 (0.14)

70. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: 12 months
Population: Echocardiogram data was available for 39 subjects in the device arm and 46 subjects in the control arm
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 39 | 46
cm^2 | 0.18 (0.12) | 0.26 (0.19)

71. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: 24 months
Population: Echocardiogram data was available for 18 subjects in the device arm and 25 subjects in the control arm
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 18 | 25
cm^2 | 0.15 (0.09) | 0.25 (0.12)

72. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: 3 years
Population: Echocardiogram data was available for 16 subjects in the device arm and 13 subjects in the control arm
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 16 | 13
cm^2 | 0.18 (0.20) | 0.18 (0.10)

73. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: 4 years
Population: Echocardiogram data was available for the 8 subjects in the device arm and 6 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 8 | 6
cm^2 | 0.14 (0.05) | 0.19 (0.12)

74. Other Pre Specified Outcome: Effective Regurgitant Orifice Area
Description: Effective Regurgitant Orifice area is defined as = Regurgitant flow / Regurgitant velocity
Time Frame: 5 years
Population: Echocardiogram data was available for the 7 subjects in the device arm and 7 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 7 | 7
cm^2 | 0.15 (0.05) | 0.15 (0.05)

75. Other Pre Specified Outcome: Regurgitant Volume
Description: Regurgitant Volume is calculated by subtracting the inflow volume across the mitral valve during diastole from the Left Ventricular Outflow Tract (LVOT) stroke volume during systole.
Time Frame: Baseline
Population: Echocardiogram data was available for 124 subjects in the device arm and 136 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 124 | 136
ml/beat | 28.80 (16.99) | 25.01 (15.31)

76. Other Pre Specified Outcome: Regurgitant Volume
Description: as for outcome 75
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: Echocardiogram data was available for 85 subjects in device arm and 70 subjects in control arm
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 85 | 70
ml/beat | 20.04 (11.86) | 25.97 (15.68)

77. Other Pre Specified Outcome: Regurgitant Volume
Description: as for outcome 75
Time Frame: 6 months
Population: Echocardiogram data was available for 45 subjects in the device arm and 54 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 45 | 54
ml/beat | 23.60 (16.00) | 32.59 (15.82)

78. Other Pre Specified Outcome: Regurgitant Volume
Description: as for outcome 75
Time Frame: 12 months
Population: Echocardiogram data was available for 33 subjects in the device arm and 45 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 33 | 45
ml/beat | 21.61 (12.12) | 27.76 (14.35)

79. Other Pre Specified Outcome: Regurgitant Volume
Description: as for outcome 75
Time Frame: 24 months
Population: Echocardiogram data was available for 21 subjects in the device arm and 28 subjects in the control arm
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 21 | 28
ml/beat | 21.48 (11.34) | 32.96 (16.04)

80. Other Pre Specified Outcome: Regurgitant Volume
Description: Regurgitant Volume is calculated by subtracting the inflow volume across the mitral valve during diastole from theLeft Ventricular Outflow Tract (LVOT) stroke volume during systole.
Time Frame: 3 years
Population: Echocardiogram data was available for 20 subjects in the device arm and 17 subjects in the control arm
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 20 | 17
ml/beat | 18.80 (9.61) | 24.65 (12.26)

81. Other Pre Specified Outcome: Regurgitant Volume
Description: as for outcome 75
Time Frame: 4 years
Population: Echocardiogram data was available for 11 subjects in the device arm and 5 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 11 | 5
ml/beat | 18.36 (6.27) | 23.00 (14.47)

82. Other Pre Specified Outcome: Regurgitant Volume
Description: as for outcome 75
Time Frame: 5 years
Population: Echocardiogram data was available for 9 subjects in the device arm and 9 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 9 | 9
ml/beat | 21.11 (10.11) | 18.78 (5.95)

83. Other Pre Specified Outcome: Regurgitant Fraction
Description: Regurgitant fraction is the percentage of blood that regurgitates back through the aortic valve to the left ventricle due to aortic insufficiency, or through the mitral valve to the atrium due to mitral insufficiency.
Time Frame: Baseline
Population: Echocardiogram data was available for 123 subjects in the device group and 136 subjects in the control group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 123 | 136
percentage | 38.24 (13.81) | 34.81 (14.94)

84. Other Pre Specified Outcome: Regurgitant Fraction
Description: as for outcome 83
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: Echocardiogram data was available for 85 subjects in the device arm and 70 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 85 | 70
percentage | 31.00 (14.53) | 35.29 (15.32)

85. Other Pre Specified Outcome: Regurgitant Fraction
Description: as for outcome 83
Time Frame: 6 months
Population: Echocardiogram data was available for 45 subjects in the device arm and 54 subjects in the control arm
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 45 | 54
percentage | 34.14 (15.89) | 42.20 (14.49)

86. Other Pre Specified Outcome: Regurgitant Fraction
Description: as for outcome 83
Time Frame: 12 months
Population: Echocardiogram data was available for 33 subjects in the device arm and 45 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 33 | 45
percentage | 32.15 (13.06) | 37.80 (15.49)

87. Other Pre Specified Outcome: Regurgitant Fraction
Description: as for outcome 83
Time Frame: 24 months
Population: Echocardiogram data is available for 21 subjects in the device arm and 28 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 21 | 28
percentage | 34.29 (14.52) | 41.79 (14.93)

88. Other Pre Specified Outcome: Regurgitant Fraction
Description: Regurgitant fraction is the percentage of blood that regurgitates back through the aortic valve to the left ventricledue to aortic insufficiency, or through the mitral valve to the atrium due to mitral insufficiency.
Time Frame: 3 years
Population: Echocardiogram data is available for 20 subjects in the device arm and 17 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 20 | 17
percentage | 31.00 (12.38) | 38.71 (10.21)

89. Other Pre Specified Outcome: Regurgitant Fraction
Description: as for outcome 83
Time Frame: 4 years
Population: Echocardiogram data was available for 11 subjects in the device arm and 5 subjects in the control arm
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 11 | 5
percentage | 32.00 (7.72) | 38.80 (21.51)

90. Other Pre Specified Outcome: Regurgitant Fraction
Description: as for outcome 83
Time Frame: 5 years
Population: Echocardiogram data is available for 9 subjects in the device arm and 9 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 9 | 9
percentage | 37.78 (12.77) | 32.78 (9.20)

91. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: Baseline
Population: All available echocardiogram data used for analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 281 | 294
mL | 194.4 (69.2) | 191.0 (72.9)

92. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 259 | 223
mL | 176.0 (64.6) | 179.1 (68.4)

93. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: 6 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 200 | 171
mL | 181.4 (65.1) | 182.6 (72.4)

94. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: 12 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 168 | 146
mL | 179.4 (66.2) | 176.3 (65.1)

95. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: 24 months
Population: All available echocardiogram data has been presented
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 121 | 94
mL | 174.5 (60.9) | 184.6 (73.5)

96. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: 3 years
Population: All available echocardiogram data has been presented
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 92 | 51
mL | 169.6 (60.5) | 172.2 (67.1)

97. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: 4 years
Population: All available electrocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 53 | 33
mL | 166.0 (58.4) | 161.6 (64.7)

98. Other Pre Specified Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricle End-diastolic volume is the amount of blood that is in the left ventricle before the heart contracts.
Time Frame: 5 years
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 37 | 32
ml | 174.0 (67.1) | 166.6 (77.0)

99. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left Ventricular End-systolic volume (LVESV) is the volume of blood in the left ventricle at the end of contraction, or systole, and the beginning of filling, or diastole. LVESV is the lowest volume of blood in the left ventricle at any point in the cardiac cycle.
Time Frame: Baseline
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 281 | 294
mL | 135.5 (56.1) | 134.3 (60.3)

100. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 99
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 258 | 223
mL | 129.3 (56.5) | 125.7 (57.1)

101. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 99
Time Frame: 6 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 200 | 171
mL | 133.1 (59.2) | 129.1 (59.2)

102. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 99
Time Frame: 12 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 168 | 146
mL | 133.0 (60.9) | 125.9 (54.8)

103. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 99
Time Frame: 24 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 121 | 94
mL | 127.4 (52.6) | 132.2 (64.7)

104. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left Ventricular End-systolic volume (LVESV) is the volume of blood in the left ventricle at the end of contraction,or systole, and the beginning of filling, or diastole. LVESV is the lowest volume of blood in the left ventricle at anypoint in the cardiac cycle.
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 92 | 51
mL | 124.3 (58.3) | 122.9 (61.1)

105. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 99
Time Frame: 4 years
Population: All available electrocardiogram has been presented.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 53 | 33
ml | 118.7 (53.1) | 112.7 (59.4)

106. Other Pre Specified Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 99
Time Frame: 5 years
Population: All available electrocardiogram has been presented.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 37 | 32
ml | 129.0 (65.4) | 119.3 (70.6)

107. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: Baseline
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 301 | 307
cm | 6.17 (0.73) | 6.19 (0.75)

108. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 286 | 249
cm | 6.10 (0.75) | 7.41 (19.58)

109. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 6 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 231 | 210
cm | 6.12 (0.77) | 6.15 (0.81)

110. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 12 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 198 | 174
cm | 6.08 (0.77) | 6.10 (0.83)

111. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 24 months
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 157 | 126
cm | 6.07 (0.92) | 6.18 (0.88)

112. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 3 years
Population: All Available echocardiogram data has been entered
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 115 | 77
cm | 6.12 (0.78) | 6.11 (0.97)

113. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 4 years
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 78 | 49
cm | 6.04 (0.81) | 6.07 (0.91)

114. Other Pre Specified Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 5 years
Population: All available echocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 57 | 45
cm | 6.09 (0.90) | 5.97 (0.91)

115. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 301 | 306
cm | 5.28 (0.86) | 5.30 (0.89)

116. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 286 | 248
cm | 5.31 (0.89) | 6.12 (12.64)

117. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 231 | 208
cm | 5.34 (0.91) | 5.28 (0.96)

118. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 197 | 173
cm | 5.26 (0.95) | 5.25 (0.99)

119. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 156 | 123
cm | 5.24 (1.07) | 5.26 (1.02)

120. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 112 | 75
cm | 5.30 (0.96) | 5.19 (1.16)

121. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 4 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 74 | 47
cm | 5.17 (0.95) | 5.01 (1.12)

122. Other Pre Specified Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 54 | 42
cm | 5.31 (1.02) | 5.15 (1.02)

123. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 281 | 294
percentage | 31.32 (9.07) | 31.30 (9.58)

124. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 259 | 223
percentage | 27.88 (8.84) | 31.11 (10.45)

125. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 200 | 171
percentage | 28.38 (10.45) | 30.44 (10.15)

126. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 168 | 146
percentage | 27.74 (11.31) | 29.72 (10.06)

127. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 121 | 94
percentage | 27.95 (9.2) | 30.68 (12.38)

128. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 92 | 51
percentage | 29.28 (12.41) | 31.67 (12.76)

129. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 4 years
Population: All available electrocardiogram has been presented.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 53 | 33
percentage | 30.87 (11.37) | 33.39 (13.09)

130. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 5 years
Population: All electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 37 | 32
percentage | 28.73 (11.26) | 32.22 (13.95)

131. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 253 | 275
mmHg | 43.95 (13.44) | 44.56 (13.96)

132. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 257 | 239
mmHg | 41.41 (11.63) | 43.81 (14.24)

133. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 196 | 188
mmHg | 40.96 (13.06) | 42.21 (14.19)

134. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 170 | 144
mmHg | 38.63 (13.00) | 39.31 (13.24)

135. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 128 | 100
mmHg | 39.46 (12.90) | 40.27 (14.92)

136. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 100 | 60
mmHg | 37.73 (11.56) | 37.57 (13.61)

137. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: 4 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 65 | 38
mmHg | 37.37 (13.04) | 39.76 (14.54)

138. Other Pre Specified Outcome: Right Ventricular Systolic Pressure (RVSP)
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 47 | 32
mmHg | 34.85 (12.92) | 35.41 (12.12)

139. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 284 | 302
cm^2 | 5.17 (1.26) | 5.16 (1.16)

140. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 174 | 235
cm^2 | 2.68 (0.92) | 4.81 (1.00)

141. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 107 | 189
cm^2 | 2.84 (1.10) | 4.94 (1.00)

142. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 106 | 142
cm^2 | 2.67 (0.86) | 4.88 (0.95)

143. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 65 | 94
cm^2 | 2.85 (1.01) | 4.98 (1.14)

144. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 48 | 39
cm^2 | 3.06 (0.90) | 4.47 (1.58)

145. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: 4 years
Population: All electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 21 | 25
cm^2 | 3.27 (0.79) | 4.39 (1.41)

146. Other Pre Specified Outcome: Mitral Valve Area
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 11 | 20
cm^2 | 3.76 (1.11) | 4.33 (1.31)

147. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: The normal area of the mitral valve orifice is about 4-6 cm2 when the mitral valve area goes below 2 cm2, the valve causes an impediment to the flow of blood into the left ventricle, creating a pressure gradient (mitral valve gradient) across the mitral valve. This gradient may increase by the rise in heart rate or cardiac output.
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 208 | 234
mmHg | 2.46 (1.05) | 2.28 (0.97)

148. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: as for outcome 147
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 282 | 184
mmHg | 4.10 (2.18) | 2.28 (1.28)

149. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: as for outcome 147
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 222 | 160
mmHg | 4.00 (1.98) | 2.28 (1.28)

150. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: as for outcome 147
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 197 | 138
mmHg | 3.88 (2.17) | 2.15 (1.30)

151. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: as for outcome 147
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 151 | 96
mmHg | 3.69 (1.76) | 2.25 (1.71)

152. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: The normal area of the mitral valve orifice is about 4-6 cm2 when the mitral valve area goes below 2 cm2, thevalve causes an impediment to the flow of blood into the left ventricle, creating a pressure gradient (mitral valvegradient) across the mitral valve. This gradient may increase by the rise in heart rate or cardiac output.
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 111 | 63
mmHg | 3.45 (1.80) | 2.62 (1.99)

153. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: as for outcome 147
Time Frame: 4 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 74 | 48
mmHg | 3.69 (1.85) | 2.56 (1.41)

154. Other Pre Specified Outcome: Mean Mitral Valve Gradient
Description: as for outcome 147
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 52 | 37
mmHg | 4.07 (2.31) | 3.54 (4.27)

155. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 300 | 310
Participants
  Present | 1 | 1
  Absent | 299 | 309

156. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 289 | 258
Participants
  Present | 1 | 1
  Absent | 288 | 257

157. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 239 | 219
Participants
  Present | 0 | 1
  Absent | 239 | 218

158. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 12 months
Population: All available echocardiogram has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 210 | 177
Participants
  Present | 0 | 0
  Absent | 210 | 177

159. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 164 | 126
Participants
  Present | 0 | 0
  Absent | 164 | 126

160. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 3 years
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 120 | 78
Participants
  Present | 0 | 0
  Absent | 120 | 78

161. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 4 years
Population: All electrocardiogram data has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 81 | 50
Participants
  Present | 0 | 0
  Absent | 81 | 50

162. Other Pre Specified Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 58 | 46
Participants
  Present | 0 | 0
  Absent | 58 | 46

163. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 238 | 251
Liters/minute | 3.61 (1.09) | 3.49 (1.08)

164. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 275 | 236
Liters/minute | 3.79 (1.17) | 3.61 (1.18)

165. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 6 months
Population: All available echocardiogram has been reported.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 217 | 199
Liters/minute | 3.53 (1.06) | 3.53 (1.16)

166. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 196 | 157
Liters/minute | 3.59 (1.07) | 3.66 (1.20)

167. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 144 | 116
Liters/minute | 3.41 (0.96) | 3.38 (1.01)

168. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 3 years
Population: All available data has been entered.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 110 | 68
L/min | 3.39 (1.01) | 3.36 (1.08)

169. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 4 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 70 | 46
liters/minute | 3.49 (0.99) | 3.42 (1.27)

170. Other Pre Specified Outcome: Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 47 | 38
liters/minute | 3.43 (1.02) | 3.41 (1.10)

171. Other Pre Specified Outcome: Forward Stroke Volume
Description: Stroke volume is the amount of blood ejected from the ventricle with each cardiac cycle. It can be readily calculated by subtracting the end-systolic volume from the end-diastolic volume.
Time Frame: Baseline
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 283 | 292
mL | 50.47 (16.52) | 50.72 (16.91)

172. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: At discharge (or 30 days if discharge echocardiogram is not available)
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 278 | 243
mL | 52.41 (17.06) | 50.75 (17.69)

173. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: 6 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 222 | 207
mL | 52.13 (16.60) | 49.89 (16.80)

174. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 200 | 165
mL | 52.33 (16.46) | 53.49 (17.73)

175. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 147 | 118
mL | 50.23 (16.02) | 49.22 (15.70)

176. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: 3 years
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 111 | 68
mL | 49.19 (15.83) | 49.42 (15.29)

177. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: 4 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 70 | 48
mL | 50.95 (16.46) | 48.32 (14.36)

178. Other Pre Specified Outcome: Forward Stroke Volume
Description: as for outcome 171
Time Frame: 5 years
Population: All available electrocardiogram data has been presented.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 47 | 38
mL | 49.70 (18.41) | 47.63 (16.75)

179. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Components of the Primary Safety Composite
Description: Freedom from the components of the primary safety composite of device related complications including Single Leaflet Device Attachment (SLDA), device embolizations, endocarditis requiring surgery, Echocardiography Core Laboratory confirmed mitral stenosis requiring surgery, LVAD implant, heart transplant, or any device related complications requiring non-elective cardiovascular surgery at 12 months will be the primary measure of safety.
Time Frame: 12 months in Device group
Population: All eligible subjects with MitraClip until the 365 day window.
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 237
percentage
  Single Leaflet Device Attachment (SLDA): number analyzed (Participants) | 236
  Single Leaflet Device Attachment (SLDA) | 99.3
  Embolization | 99.7
  Left Ventricular Assist Device (LVAD): number analyzed (Participants) | 235
  Left Ventricular Assist Device (LVAD) | 98.8
  Heart Transplant: number analyzed (Participants) | 235
  Heart Transplant | 99.2
  Non-elective Cardiovascular surgery | 99.7

180. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Components of the Primary Safety Composite
Description: as for outcome 179
Time Frame: 24 months in Device group
Population: All available subjects with data within the 2 year (731 days) window
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 204
percentage
  Single Leaflet Device Attachment (SLDA): number analyzed (Participants) | 203
  Single Leaflet Device Attachment (SLDA) | 99.3
  Embolization | 99.7
  Left Ventricular Assist Device (LVAD): number analyzed (Participants) | 201
  Left Ventricular Assist Device (LVAD) | 97.4
  Heart Transplant: number analyzed (Participants) | 201
  Heart Transplant | 98.7
  Non-elective cardiovascular surgery | 99.7

181. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Components of the Primary Safety Composite
Description: as for outcome 179
Time Frame: 3 years in Device group
Population: All available subjects within the 36 month (1096 days) window.
Measure: Number; unit: Percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 164
Percentage
  Single Leaflet DeviceAttachment (SLDA) | 99.3
  Embolization | 99.7
  Left Ventricular AssistDevice (LVAD): number analyzed (Participants) | 159
  Left Ventricular AssistDevice (LVAD) | 94.9
  Heart Transplant: number analyzed (Participants) | 158
  Heart Transplant | 96.6
  Non-electivecardiovascular surgery | 99.7

182. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Components of the Primary Safety Composite
Description: Freedom from the components of the primary safety composite of device relatedcomplications including Single Leaflet Device Attachment (SLDA), deviceembolizations, endocarditis requiring surgery, Echocardiography Core Laboratoryconfirmed mitral stenosis requiring surgery, LVAD implant, heart transplant, or any device related complications requiring non-elective cardiovascular surgery at12 months will be the primary measure of safety.
Time Frame: 4 years in Device group
Population: All subjects within the 4 year (1461 days) window.
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 138
percentage
  Single Leaflet Device Attachment (SLDA) | 99.3
  Embolization | 99.7
  Left Ventricular Assist Device (LVAD): number analyzed (Participants) | 134
  Left Ventricular Assist Device (LVAD) | 94.2
  Heart Transplant: number analyzed (Participants) | 131
  Heart Transplant | 95.3
  Non-elective Cardiovascular Surgery | 99.7

183. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Components of the Primary Safety Composite
Description: Freedom from the components of the primary safety composite of device related complications including Single Leaflet Device Attachment (SLDA), device embolizations, endocarditis requiring surgery, Echocardiography Core Laboratory confirmed mitral stenosis requiring surgery, LVAD implant, heart transplant, or any device related complications requiring non-elective cardiovascular surgery at12 months will be the primary measure of safety.
Time Frame: 5 years in Device group
Population: All available subjects within 5 year (1826 days) window.
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 70
percentage
  Single LeafletDeviceAttachment(SLDA) | 99.3
  Embolization | 99.7
  Left VentricularAssistDevice (LVAD): number analyzed (Participants) | 66
  Left VentricularAssistDevice (LVAD) | 93.5
  Heart Transplant: number analyzed (Participants) | 65
  Heart Transplant | 95.3
  Non-electivecardiovascularsurgery | 99.7

184. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Primary Safety Composite
Description: Freedom from the primary safety composite of device related complications including Single Leaflet Device Attachment (SLDA), device embolizations, endocarditis requiring surgery, Echocardiography Core Laboratory confirmed mitral stenosis requiring surgery, LVAD implant, heart transplant, or any device related complications requiring non-elective cardiovascular surgery at 12 months will be the primary measure of safety.
Time Frame: 24 months in Device group
Population: All available subjects with data within the 24 months (731 days) window.
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 197
percentage | 94.8

185. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Primary Safety Composite
Description: Freedom from the primary safety composite of device related complications including Single Leaflet DeviceAttachment (SLDA), device embolizations, endocarditis requiring surgery, Echocardiography Core Laboratoryconfirmed mitral stenosis requiring surgery, LVAD implant, heart transplant, or any device related complicationsrequiring non-elective cardiovascular surgery at 12 months will be the primary measure of safety.
Time Frame: 3 years in Device group
Population: All available subjects with data within the 36 months (1096 days) window.
Measure: Number; unit: Percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 154
Percentage | 91.2

186. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Primary Safety Composite
Description: as for outcome 184
Time Frame: 4 years in Device group
Population: All available echocardiogram data has been presented.
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 128
percentage | 89.9

187. Other Pre Specified Outcome: Kaplan-Meier Freedom From the Primary Safety Composite
Description: as for outcome 184
Time Frame: 5 years in Device group
Population: All available electrocardiogram has been presented.
Measure: Number; unit: percentage
Arm/Group | MitraClip System
Number analyzed (Participants) | 62
percentage | 89.2

188. Other Pre Specified Outcome: Kaplan-Meier Freedom From All-cause Mortality
Description: Kaplan-Meier survival rate for all cause mortality at 24 months
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 205 | 157
percentage | 71.9 [66.4 to 76.6] | 57.3 [51.4 to 62.8]

189. Other Pre Specified Outcome: Kaplan-Meier Freedom From All-cause Mortality
Description: Kaplan-Meier survival rate for all cause mortality at 36 months
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 167 | 122
Percentage | 59.7 [53.8 to 65.1] | 45.9 [40.0 to 51.6]

190. Other Pre Specified Outcome: Kaplan-Meier Freedom From All-cause Mortality
Description: Kaplan-Meier survival rate for all cause mortality at 48 months
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 138 | 94
percentage | 51.3 [45.4 to 57.0] | 37.3 [31.6 to 43.0]

191. Other Pre Specified Outcome: Kaplan-Meier Freedom From All-cause Mortality
Description: Kaplan-Meier survival rate for all cause mortality at 60 months
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 79 | 59
percentage | 42.7 [36.8 to 48.5] | 32.8 [27.2 to 38.4]

192. Other Pre Specified Outcome: Kaplan-Meier Freedom From Cardiovascular Mortality
Description: Kaplan-Meier survival rate for Cardiovascular mortality.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 238 | 223
percentage | 86.2 [81.6 to 89.7] | 80.7 [75.7 to 84.8]

193. Other Pre Specified Outcome: Kaplan-Meier Freedom From Cardiovascular Mortality
Description: Kaplan-Meier survival rate for Cardiovascular mortality.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 205 | 156
percentage | 77.6 [72.3 to 82.1] | 64.5 [58.6 to 69.9]

194. Other Pre Specified Outcome: Kaplan-Meier Freedom From Cardiovascular Mortality
Description: Kaplan-Meier survival rate for Cardiovascular mortality.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 167 | 120
Percentage | 66.7 [60.7 to 72.0] | 54.6 [48.3 to 60.5]

195. Other Pre Specified Outcome: Kaplan-Meier Freedom From Cardiovascular Mortality
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 138 | 94
percentage | 58.8 [52.6 to 64.5] | 47.0 [40.6 to 53.1]

196. Other Pre Specified Outcome: Kaplan-Meier Freedom From Cardiovascular Mortality
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 79 | 59
percentage | 51.2 [44.8 to 57.2] | 42.8 [36.4 to 49.0]

197. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 194 | 157
Percentage | 74.4 [68.9 to 79.1] | 60.4 [54.5 to 65.7]

198. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 158 | 95
Percentage | 64.5 [58.5 to 69.9] | 43.9 [37.9 to 49.8]

199. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 118 | 43
Percentage | 53.2 [46.9 to 59.2] | 23.6 [18.2 to 29.3]

200. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 93 | 33
percentage | 45.7 [39.3 to 51.8] | 22.3 [17.0 to 28.1]

201. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 52 | 17
percentage | 39.0 [32.6 to 45.4] | 17.0 [11.9 to 22.8]

202. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First Cardiovascular Hospitalization
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 166 | 137
Percentage | 61.7 [55.8 to 67.1] | 51.3 [45.5 to 56.9]

203. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First Cardiovascular Hospitalization
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 126 | 78
Percentage | 49.5 [43.5 to 55.2] | 33.5 [27.9 to 39.2]

204. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First Cardiovascular Hospitalization
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 87 | 36
Percentage | 37.3 [31.4 to 43.1] | 17.5 [12.9 to 22.6]

205. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First Cardiovascular Hospitalization
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 63 | 26
Percentage | 28.5 [23.0 to 34.2] | 14.8 [10.5 to 19.8]

206. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First Cardiovascular Hospitalization
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 34 | 11
Percentage | 23.0 [17.9 to 28.6] | 10.8 [7.0 to 15.6]

207. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization or All-cause Mortality
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 196 | 156
Percentage | 66.5 [60.8 to 71.5] | 53.8 [48.1 to 59.2]

208. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization or All-cause Mortality
Description: Survival rate from the first HF related hospitalization or all-cause mortality.
Time Frame: 24 months
Population: All available data has been reported.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 158 | 95
percentage | 54.8 [48.9 to 60.3] | 33.8 [28.4 to 39.2]

209. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization or All-cause Mortality
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 118 | 43
Percentage | 41.5 [35.8 to 47.1] | 15.5 [11.5 to 20.0]

210. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization or All-cause Mortality
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 93 | 33
percentage | 34.0 [28.6 to 39.5] | 12.8 [9.1 to 17.0]

211. Other Pre Specified Outcome: Kaplan-Meier Freedom From the First HF Related Hospitalization or All-cause Mortality
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 52 | 17
percentage | 26.4 [21.4 to 31.7] | 8.5 [5.5 to 12.3]

212. Other Pre Specified Outcome: NYHA Functional Class
Description: Measure Description: The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity:
  Class I: No symptoms and no limitation in ordinary physical activity Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity Class III: Marked limitation in activity due to symptoms Class IV: Severe limitations
Time Frame: Baseline
Population: NYHA Class data available for only 311 subjects
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  NYHA Class I: number analyzed (Participants) | 302 | 311
  NYHA Class I | 1 | 0
  NYHA Class II: number analyzed (Participants) | 302 | 311
  NYHA Class II | 129 | 110
  NYHA Class III: number analyzed (Participants) | 302 | 311
  NYHA Class III | 154 | 168
  NYHA Class IV: number analyzed (Participants) | 302 | 311
  NYHA Class IV | 18 | 33

213. Other Pre Specified Outcome: NYHA Functional Class
Description: as for outcome 212
Time Frame: 30 days
Population: All available data at 30 day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 281 | 278
Participants
  NYHA Class I | 44 | 14
  NYHA Class II | 172 | 120
  NYHA Class III | 55 | 117
  NYHA Class IV | 10 | 27

214. Other Pre Specified Outcome: NYHA Functional Class
Description: as for outcome 212
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 253 | 238
Participants
  NYHA Class I | 51 | 14
  NYHA Class II | 139 | 117
  NYHA Class III | 56 | 100
  NYHA Class IV | 7 | 7

215. Other Pre Specified Outcome: NYHA Functional Class
Description: as for outcome 212
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 219 | 191
Participants
  NYHA Class I | 40 | 18
  NYHA Class II | 131 | 97
  NYHA Class III | 42 | 65
  NYHA Class IV | 6 | 11

216. Other Pre Specified Outcome: NYHA Functional Class
Description: as for outcome 212
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 176 | 143
Participants
  NYHA Class I | 31 | 12
  NYHA Class II | 91 | 69
  NYHA Class III | 44 | 54
  NYHA Class IV | 10 | 8

217. Other Pre Specified Outcome: NYHA Functional Class
Description: Measure Description: The New York Heart Association (NYHA) Classification provides a simple way of classifyingthe extent of heart failure. It classifies patients in one of four categories based on their limitations during physicalactivity:
  Class I: No symptoms and no limitation in ordinary physical activity Class II: Mild symptoms (mild shortness ofbreath and/or angina) and slight limitation during ordinary activity Class III: Marked limitation in activity due tosymptoms Class IV: Severe limitations
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 146 | 102
Participants
  NYHA Class I | 25 | 16
  NYHA Class II | 85 | 48
  NYHA Class III | 32 | 32
  NYHA Class IV | 4 | 6

218. Other Pre Specified Outcome: NYHA Functional Class
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 125 | 76
Participants
  NYHA Class I | 21 | 10
  NYHA Class II | 70 | 36
  NYHA Class III | 29 | 25
  NYHA Class IV | 5 | 5

219. Other Pre Specified Outcome: NYHA Functional Class
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 94 | 65
Participants
  NYHA Class I | 17 | 12
  NYHA Class II | 45 | 27
  NYHA Class III | 28 | 26
  NYHA Class IV | 4 | 0

220. Other Pre Specified Outcome: Six-Minute Walk Test Distance (6MWD)
Description: Six-Minute Walk Test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk test distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Time Frame: Baseline
Population: All available 6MWD has been reported.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 296 | 305
meters | 249.6 (123.8) | 234.5 (123.5)

221. Other Pre Specified Outcome: 6MWD
Description: as for outcome 220
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 265 | 244
meters | 290.1 (122.8) | 243.0 (121.0)

222. Other Pre Specified Outcome: 6MWD
Description: as for outcome 220
Time Frame: 6 months
Population: All available 6MWD has been reported
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 237 | 203
meters | 288.6 (128.0) | 253.9 (126.2)

223. Other Pre Specified Outcome: 6MWD
Description: as for outcome 220
Time Frame: 12 months
Population: All available 6MWD has been reported
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 193 | 167
meters | 308.4 (116.7) | 269.7 (133.2)

224. Other Pre Specified Outcome: 6MWD
Description: as for outcome 220
Time Frame: 24 months
Population: All available 6MWD has been reported.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 143 | 111
meters | 294.2 (131.2) | 273.8 (142.7)

225. Other Pre Specified Outcome: Change in 6MWD From Baseline
Time Frame: Between baseline and 30 days
Population: All available data has been reported
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 260 | 243
meters | 31.6 (106.4) | -0.9 (83.5)

226. Other Pre Specified Outcome: Change in 6MWD From Baseline
Time Frame: Between baseline and 6 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 233 | 201
meters | 25.9 (100.6) | 0.66 (99.9)

227. Other Pre Specified Outcome: Change in 6MWD From Baseline
Time Frame: Between baseline and 12 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 191 | 166
meters | 33.9 (99.6) | 5.5 (115.0)

228. Other Pre Specified Outcome: Change in 6MWD From Baseline
Time Frame: Between baseline and 24 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 142 | 110
meters | 12.5 (103.0) | 1.1 (133.6)

229. Other Pre Specified Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) QoL Scores
Description: The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score.
  Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification.
  Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: Baseline
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 309
KCCQ score on a points scale | 53.2 (22.8) | 51.6 (23.3)

230. Other Pre Specified Outcome: KCCQ QoL Scores
Description: as for outcome 229
Time Frame: 30 days
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 279 | 275
KCCQ score on a points scale | 70.9 (21.1) | 54.6 (24.7)

231. Other Pre Specified Outcome: KCCQ QoL Scores
Description: as for outcome 229
Time Frame: 6 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 252 | 237
KCCQ score on a points scale | 73.0 (21.3) | 59.0 (24.7)

232. Other Pre Specified Outcome: KCCQ QoL Scores
Description: as for outcome 229
Time Frame: 12 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 219 | 189
KCCQ score on a points scale | 71.8 (22.2) | 60.2 (24.5)

233. Other Pre Specified Outcome: KCCQ QoL Scores
Description: as for outcome 229
Time Frame: 24 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 175 | 138
KCCQ score on a points scale | 71.3 (23.3) | 58.9 (25.2)

234. Other Pre Specified Outcome: Change in KCCQ QoL Scores From Baseline
Description: Paired data looking at difference between the baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) and 30 days KCCQ score.
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score.
  Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification.
  Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: Between baseline and 30 days
Population: All available paired data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 279 | 272
KCCQ score on a points scale | 16.9 (22.8) | 2.1 (18.6)

235. Other Pre Specified Outcome: Change in KCCQ QoL Scores From Baseline
Description: Paired data looking at difference between the baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) and 6 months KCCQ score.
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score.
  Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification.
  Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: Between baseline and 6 months
Population: All available paired data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 252 | 236
KCCQ score on a points scale | 18.5 (24.9) | 5.3 (23.0)

236. Other Pre Specified Outcome: Change in KCCQ QoL Scores From Baseline
Description: Paired data looking at difference between the baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) and 12 months KCCQ score.
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score.
  Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification.
  Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: Between baseline and 12 months
Population: All available paired data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 219 | 188
KCCQ score on a points scale | 17.0 (25.4) | 5.1 (24.5)

237. Other Pre Specified Outcome: Change in KCCQ QoL Scores From Baseline
Description: Paired data looking at difference between the baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) and 24 months KCCQ score.
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score.
  Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification.
  Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.
Time Frame: Between baseline and 24 months
Population: All available paired data has been reported.
Measure: Mean (Standard Deviation); unit: KCCQ score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 175 | 138
KCCQ score on a points scale | 17.4 (25.8) | 3.4 (26.5)

238. Other Pre Specified Outcome: SF-36 QoL Scores
Description: The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Time Frame: Baseline
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 299 | 308
SF-36 score on a points scale
  SF-36 PCS | 33.0 (9.1) | 32.6 (10.0)
  SF-36 MCS | 46.7 (12.7) | 13.0 (12.0)

239. Other Pre Specified Outcome: SF-36 QoL Scores
Description: as for outcome 238
Time Frame: 30 days
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 278 | 272
SF-36 score on a points scale
  SF-36 PCS | 39.2 (9.2) | 33.6 (9.9)
  SF-36 MCS | 51.4 (11.5) | 46.1 (13.4)

240. Other Pre Specified Outcome: SF-36 QoL Scores
Description: as for outcome 238
Time Frame: 6 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 scores on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 251 | 237
SF-36 scores on a points scale
  SF-36 PCS | 39.0 (10.3) | 34.2 (9.9)
  SF-36 MCS | 52.1 (10.3) | 47.0 (12.9)

241. Other Pre Specified Outcome: SF-36 QoL Scores
Description: as for outcome 238
Time Frame: 12 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 scores on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 218 | 190
SF-36 scores on a points scale
  SF-36 PCS | 38.7 (10.2) | 34.6 (10.8)
  SF-36 MCS | 51.3 (10.8) | 48.2 (13.8)

242. Other Pre Specified Outcome: SF-36 QoL Scores
Description: as for outcome 238
Time Frame: 24 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 scores on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 174 | 137
SF-36 scores on a points scale
  SF-36 PCS | 38.7 (10.4) | 33.7 (9.8)
  SF-36 MCS | 50.6 (12.1) | 47.2 (12.1)

243. Other Pre Specified Outcome: Change in SF-36 QoL Scores From Baseline
Description: Paired data looking at difference between the baseline SF-36 and 30 days SF-36. The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Time Frame: Between baseline and 30 days
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 276 | 269
SF-36 score on a points scale
  SF-36 PCS | 6.0 (8.9) | 0.6 (8.1)
  SF_36 MCS | 4.2 (12.2) | 0.4 (12.0)

244. Other Pre Specified Outcome: Change in SF-36 QoL Scores From Baseline
Description: Paired data looking at difference between the baseline SF-36 and 6 months days SF-36.
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Time Frame: Between baseline and 6 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 248 | 234
SF-36 score on a points scale
  SF-36 PCS | 5.5 (10.2) | 1.0 (8.7)
  SF-36 MCS | 4.6 (12.2) | 1.1 (10.7)

245. Other Pre Specified Outcome: Change in SF-36 QoL Scores From Baseline
Description: Paired data looking at difference between the baseline SF-36 and 12 month SF-36.
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Time Frame: Between baseline and 12 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 215 | 187
SF-36 score on a points scale
  SF-36 PCS | 5.0 (10.4) | 0.8 (9.8)
  SF-36 MCS | 4.3 (13.2) | 1.9 (13.4)

246. Other Pre Specified Outcome: Change in SF-36 QoL Scores From Baseline
Description: Paired data looking at difference between the baseline SF-36 and 24 months SF-36.
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Time Frame: Between baseline and 24 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: SF-36 score on a points scale
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 171 | 136
SF-36 score on a points scale
  SF-36 PCS | 5.0 (10.4) | 0.7 (10.6)
  SF-36 MCS | 3.8 (14.2) | -0.3 (12.9)

247. Other Pre Specified Outcome: Mitral Valve Surgery (Including Type of Surgery), New Use of CRT, New Use of Single or Dual Chamber Pacemaker, Permanent LVAD Implant, Heart Transplant, Additional MitraClip Device Intervention in Device Group
Time Frame: Through 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  Mitral Valve Surgery Elective - Repair | 0 | 3
  Mitral Valve Surgery Elective - Replacement | 1 | 5
  Mitral Valve Surgery Non Elective - Repair | 0 | 0
  Mitral Valve Surgery Non Elective - Replacement | 0 | 0
  New Use of CRT | 8 | 11
  New use of single or dual chamber Pacemaker | 10 | 10
  Permanent LVAD Implant | 16 | 18
  Heart Transplant | 9 | 11
  Additional MitraClip Device Intervention | 10 | NA — MitraClip Intervention is not applicable for Control Group

248. Other Pre Specified Outcome: De Novo MitraClip Device Intervention in Control Group
Time Frame: Through 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | NA — This is only applicable for Control Group | 67

249. Other Pre Specified Outcome: Responder Analysis for 6MWD
Description: Where responder is defined as alive and experiencing an improvement of 24 meters and 50 meters (difference in proportion of responders between Device and Control groups)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 191 | 166
Participants
  Experiencing Improvement >= 24 meters | 100 | 66
  Experiencing Improvement >= 50 meters | 75 | 42

250. Other Pre Specified Outcome: Responder Analysis for 6MWD
Description: as for outcome 249
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 106 | 72
Participants
  Experiencing Improvement >= 24 meters | 44 | 34
  Experiencing Improvement >= 50 meters | 34 | 23

251. Other Pre Specified Outcome: Responder Analysis for LVEDV Index
Description: Where responder is defined as alive and experiencing an improvement of 12 ml/m2 (difference in proportion of responders between Device and Control groups)
Time Frame: 12 months
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 160 | 130
Participants | 35 | 32

252. Other Pre Specified Outcome: Responder Analysis for LVEDV Index
Description: as for outcome 251
Time Frame: 24 months
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 115 | 89
Participants | 26 | 20

253. Other Pre Specified Outcome: Responder Analysis for LVEDV Index
Description: as for outcome 251
Time Frame: 3 years
Population: All available echocardiogram data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 88 | 43
Participants | 20 | 8

254. Other Pre Specified Outcome: Responder Analysis for LVEDV Index
Description: as for outcome 251
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 53 | 28
Participants | 13 | 6

255. Other Pre Specified Outcome: Responder Analysis for LVEDV Index
Description: as for outcome 251
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 36 | 26
Participants | 9 | 3

256. Other Pre Specified Outcome: Responder Analysis for QoL (KCCQ)
Description: Where responder is defined as alive and experiencing an improvement of 5 points (difference in proportion of responders between Device and Control groups)
Time Frame: 12 months
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 219 | 188
Participants | 151 | 103

257. Other Pre Specified Outcome: Responder Analysis for QoL (KCCQ)
Description: as for outcome 256
Time Frame: 24 months
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 128 | 90
Participants | 88 | 46

258. Other Pre Specified Outcome: Each Subscale for QoL (KCCQ)
Description: difference in means between Device and Control groups for the Kansas City Cardiomyopathy Questionnaire (KCCQ) for the physical limitation and symptom stability scores.
Time Frame: 12 months
Population: 219 subjects from device group and 189 subjects from control group analyzed.
Measure: Number (95% Confidence Interval); unit: KCCQ score on a points scale
Arm/Group | Randomized Group
Number analyzed (Participants) | 408
KCCQ score on a points scale | 9.90 [5.51 to 14.29]

259. Other Pre Specified Outcome: Each Subscale for QoL (KCCQ)
Description: as for outcome 258
Time Frame: 24 months
Population: 128 subjects in the device group and 90 subjects in the control group were analyzed.
Measure: Number (95% Confidence Interval); unit: KCCQ score on a points scale
Arm/Group | Randomized Group
Number analyzed (Participants) | 218
KCCQ score on a points scale | 8.01 [1.68 to 14.35]

260. Other Pre Specified Outcome: Length of Index Hospitalization for MitraClip Procedure (Device Group)
Description: Length of stay in the hospital for the MitraClip Index procedure (device group)
Time Frame: Before MitraClip procedure on day 0
Population: Data was available for 293 subjects out of 302 subjects in the device group.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MitraClip System
Number analyzed (Participants) | 293
Days | 2.5 (2.3)

261. Other Pre Specified Outcome: Number of Hospitalizations and Reason for Hospitalization (i.e. Heart Failure, Cardiovascular, Non-cardiovascular)
Description: in each of the Device and Control groups
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  Heart Failure | 70 | 118
  Cardiovascular | 52 | 54
  Non-Cardiovascular | 95 | 97

262. Other Pre Specified Outcome: Number of Hospitalizations and Reason for Hospitalization (i.e. Heart Failure, Cardiovascular, Non-cardiovascular)
Description: in each of the Device and Control groups
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  Heart Failure | 92 | 151
  Cardiovascular | 72 | 72
  Non-Cardiovascular | 124 | 128

263. Other Pre Specified Outcome: Number of Days Alive and Out of Hospital
Description: mean no of days alive and out of hospital in both Device and Control groups
Time Frame: From the time of randomization to 12 months
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of days | 316.6 (93.9) | 305.4 (98.6)

264. Other Pre Specified Outcome: Number of Days Alive and Out of Hospital
Description: mean Number of days alive and out of hospital for the Device and Control groups
Time Frame: From the time of randomization to 24 months
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 579.4 (234.0) | 521.1 (245)

265. Other Pre Specified Outcome: Number of Days Alive and Out of Hospital
Description: Mean Number of days alive and out of hospital for the Device and Control groups
Time Frame: From the time of randomization to 3 Years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 799.0 (380.9) | 676.6 (389.9)

266. Other Pre Specified Outcome: Number of Days Alive and Out of Hospital
Description: difference in medians between Device and Control groups
Time Frame: From the time of randomization to 4 Years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 979.3 (527.4) | 797.5 (527.4)

267. Other Pre Specified Outcome: Number of Days Alive and Out of Hospital
Description: difference in medians between Device and Control groups
Time Frame: From the time of randomization to 5 Years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 1123.5 (664.8) | 894.8 (655.1)

268. Other Pre Specified Outcome: Number of Days Hospitalized From the "Treatment" Visit
Description: mean Number of days hospitalized from the "Treatment" visit for the Device and Control groups
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 9.2 (14.7) | 9.6 (16.9)

269. Other Pre Specified Outcome: Number of Days Hospitalized From the "Treatment" Visit
Description: mean Number of days hospitalized from the "Treatment" visit for the Device and Control groups
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 13.0 (20.0) | 13.9 (19.8)

270. Other Pre Specified Outcome: Number of Days Hospitalized From the "Treatment" Visit
Description: mean Number of days hospitalized from the "Treatment" visit for the Device and Control groups
Time Frame: 3 Years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 18.4 (28.3) | 17.5 (22.7)

271. Other Pre Specified Outcome: Number of Days Hospitalized From the "Treatment" Visit
Description: difference in medians between Device and Control groups
Time Frame: 4 Years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 21.3 (31.1) | 19.0 (23.9)

272. Other Pre Specified Outcome: Number of Days Hospitalized From the "Treatment" Visit
Description: difference in medians between Device and Control groups
Time Frame: 5 Years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 23.8 (33.7) | 19.8 (24.1)

273. Other Pre Specified Outcome: Proportion of Alive Time in Hospital
Description: summarized and compared between Device and Control groups
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 0.05 (0.10) | 0.04 (0.09)

274. Other Pre Specified Outcome: Proportion of Alive Time in Hospital
Description: summarized and compared between Device and Control groups
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Number of Days | 0.04 (0.10) | 0.04 (0.08)

275. Other Pre Specified Outcome: Proportion of Alive Time in Hospital
Description: summarized and compared between Device and Control groups
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 311
Number of Days | 0.05 (0.10) | 0.05 (0.08)

276. Other Pre Specified Outcome: Proportion of Alive Time in Hospital
Description: summarized and compared between Device and Control groups
Time Frame: 4 years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 311
Number of Days | 0.05 (0.10) | 0.05 (0.08)

277. Other Pre Specified Outcome: Proportion of Alive Time in Hospital
Description: summarized and compared between Device and Control groups
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 311
Number of Days | 0.05 (0.10) | 0.05 (0.08)

278. Other Pre Specified Outcome: Proportion of Subjects Living in the Baseline Location
Description: Subjects living in the baseline location include : home, retirement home, nursing facility and other location.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 223 | 206
Participants | 217 | 198

279. Other Pre Specified Outcome: Proportion of Subjects Living in the Baseline Location
Description: Subjects living in the baseline location include : home, retirement home, nursing facility and other location.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 132 | 93
Participants | 130 | 87

280. Other Pre Specified Outcome: Proportion of Subjects Living in the Baseline Location
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 154 | 113
Participants | 150 | 108

281. Other Pre Specified Outcome: Proportion of Subjects Living in the Baseline Location
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 132 | 89
Participants | 129 | 86

282. Other Pre Specified Outcome: Proportion of Subjects Living in the Baseline Location
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 107 | 78
Participants | 98 | 72

283. Other Pre Specified Outcome: Mitral Valve Replacement Rates
Description: Subjects with mitral valve replacements in the Device and Control groups
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 1 | 5

284. Other Pre Specified Outcome: Mitral Valve Replacement Rates
Description: Subjects with mitral valve replacements in the Device and Control groups
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 1 | 5

285. Other Pre Specified Outcome: Mitral Valve Replacement Rates
Description: summarized and compared between Device and Control groups
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 1 | 5

286. Other Pre Specified Outcome: Mitral Valve Replacement Rates
Description: summarized and compared between Device and Control groups
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 1 | 5

287. Other Pre Specified Outcome: Mitral Valve Replacement Rates
Description: summarized and compared between Device and Control groups
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 1 | 5

288. Other Pre Specified Outcome: New Onset of Permanent Atrial Fibrillation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 14 | 13

289. Other Pre Specified Outcome: New Onset of Permanent Atrial Fibrillation
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 18 | 15

290. Other Pre Specified Outcome: New Onset of Permanent Atrial Fibrillation
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 22 | 20

291. Other Pre Specified Outcome: New Onset of Permanent Atrial Fibrillation
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 23 | 20

292. Other Pre Specified Outcome: New Onset of Permanent Atrial Fibrillation
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 23 | 23

293. Other Pre Specified Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice area of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 18 | 1

294. Other Pre Specified Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice area of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 25 | 0

295. Other Pre Specified Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice area of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 22 | 1

296. Other Pre Specified Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice area of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 23 | 2

297. Other Pre Specified Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice area of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 23 | 0

298. Other Pre Specified Outcome: Clinically Significant Atrial Septal Defect (ASD) That Requires Intervention
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 2 | 0

299. Other Pre Specified Outcome: Clinically Significant Atrial Septal Defect (ASD) That Requires Intervention
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 2 | 0

300. Other Pre Specified Outcome: Clinically Significant Atrial Septal Defect (ASD) That Requires Intervention
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 2 | 0

301. Other Pre Specified Outcome: Clinically Significant Atrial Septal Defect (ASD) That Requires Intervention
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 2 | 0

302. Other Pre Specified Outcome: Clinically Significant Atrial Septal Defect (ASD) That Requires Intervention
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 2 | 0

303. Other Pre Specified Outcome: Device-related Complications in Device Group Subjects and Control Group Subjects Who Undergo the MitraClip Procedure
Time Frame: Through 5 years
Reporting Status: Not Posted

304. Other Pre Specified Outcome: Brain Natriuretic Peptide (BNP) or N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP Levels)
Time Frame: Baseline
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
pg/ml
  BNP: number analyzed (Participants) | 208 | 209
  BNP | 1014.77 (1085.98) | 1017.13 (1212.77)
  NT-proBNP: number analyzed (Participants) | 74 | 85
  NT-proBNP | 5174.33 (6566.61) | 5943.86 (8437.61)

305. Other Pre Specified Outcome: BNP or NT-proBNP Levels
Time Frame: 30 days
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
pg/ml
  BNP: number analyzed (Participants) | 193 | 188
  BNP | 875.91 (931.18) | 1065.55 (1206.34)
  NT-proBNP: number analyzed (Participants) | 74 | 77
  NT-proBNP | 4907.58 (7483.72) | 5244.16 (7851.05)

306. Other Pre Specified Outcome: BNP or NT-proBNP Levels
Time Frame: 12 months
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
pg/ml
  BNP: number analyzed (Participants) | 146 | 122
  BNP | 621.45 (606.99) | 808.26 (1711.71)
  NT-proBNP: number analyzed (Participants) | 63 | 61
  NT-proBNP | 3362.49 (4332.12) | 3977.80 (5689.70)

307. Other Pre Specified Outcome: Modified Rankin Scale Score
Description: MODIFIED RANKIN SCALE SCORE DESCRIPTIONS:
  0- No symptoms at all; 1- No significant disability despite symptoms; able to carry out all usual duties and activities; 2- Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance; 3- Moderate disability; requiring some help, but able to walk without assistance; 4- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5- Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6- Dead
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 308
Participants
  0 | 170 | 158
  1 | 52 | 55
  2 | 55 | 58
  3 | 23 | 35
  4 | 2 | 2
  5 | 0 | 0

308. Other Pre Specified Outcome: Modified Rankin Scale Score
Description: as for outcome 307
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 278 | 276
Participants
  0 | 169 | 129
  1 | 56 | 54
  2 | 40 | 49
  3 | 13 | 34
  4 | 0 | 8
  5 | 0 | 2

309. Other Pre Specified Outcome: Modified Rankin Scale Score
Description: as for outcome 307
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 250 | 234
Participants
  0 | 145 | 120
  1 | 60 | 48
  2 | 30 | 38
  3 | 13 | 20
  4 | 2 | 8
  5 | 0 | 0

310. Other Pre Specified Outcome: Modified Rankin Scale Score
Description: as for outcome 307
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 219 | 189
Participants
  0 | 134 | 100
  1 | 42 | 40
  2 | 34 | 27
  3 | 9 | 14
  4 | 0 | 7
  5 | 0 | 1

311. Other Pre Specified Outcome: Major Bleeding
Description: Major bleeding is defined as bleeding ≥ Type 3 based on a modified Bleeding Academic Research Consortium (BARC) definition
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants | 15 | 3

312. Other Pre Specified Outcome: Prolonged Ventilation
Description: Defined as pulmonary insufficiency requiring ventilatory support for greater than 48 hours post-catheterization
Time Frame: 30 days
Reporting Status: Not Posted

313. Other Pre Specified Outcome: Average Dosages of Guideline Directed Medical Therapy (GDMT)
Time Frame: Baseline
Population: All available data has been reported and includes subjects on the drugs mentioned below. Not all subjects were on all the drugs.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE Inhibitors: number analyzed (Participants) | 138 | 115
  ACE Inhibitors | 14.18 (15.19) | 13.44 (13.56)
  Angiotensin-Receptor Blockers (ARB): number analyzed (Participants) | 66 | 71
  Angiotensin-Receptor Blockers (ARB) | 14.21 (9.37) | 12.35 (8.69)
  Aldosterone Antagonists: number analyzed (Participants) | 153 | 154
  Aldosterone Antagonists | 24.51 (11.62) | 28.96 (34.12)
  Beta Blockers: number analyzed (Participants) | 275 | 278
  Beta Blockers | 31.91 (24.90) | 29.92 (25.79)
  Vasodilators (Nitrate): number analyzed (Participants) | 19 | 25
  Vasodilators (Nitrate) | 59.61 (43.81) | 42.80 (26.97)
  Vasodilators (Hydralazine): number analyzed (Participants) | 50 | 55
  Vasodilators (Hydralazine) | 139.85 (108.46) | 109.27 (86.45)
  ARN Inhibitors: number analyzed (Participants) | 13 | 9
  ARN Inhibitors | 12.64 (9.31) | 9.65 (6.80)

314. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 30 days
Population: as for outcome 313
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE Inhibitors: number analyzed (Participants) | 138 | 115
  ACE Inhibitors | 13.61 (15.01) | 13.53 (13.68)
  Angiotensin Receptor Blockers (ARBs): number analyzed (Participants) | 65 | 75
  Angiotensin Receptor Blockers (ARBs) | 13.68 (9.34) | 11.89 (8.76)
  Aldosterone Antagonists: number analyzed (Participants) | 154 | 154
  Aldosterone Antagonists | 24.21 (11.56) | 29.48 (34.36)
  Beta Blockers: number analyzed (Participants) | 278 | 281
  Beta Blockers | 30.12 (24.81) | 29.25 (25.26)
  Vasodilators (Nitrate): number analyzed (Participants) | 21 | 29
  Vasodilators (Nitrate) | 56.38 (42.76) | 43.79 (27.15)
  Vasodilators (Hydralazine): number analyzed (Participants) | 51 | 57
  Vasodilators (Hydralazine) | 133.41 (108.29) | 110.53 (87.72)
  ARN Inhibitors: number analyzed (Participants) | 15 | 12
  ARN Inhibitors | 13.17 (11.15) | 8.85 (5.98)

315. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 6 months
Population: as for outcome 313
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE I: number analyzed (Participants) | 143 | 116
  ACE I | 13.22 (14.59) | 12.90 (12.96)
  ARB: number analyzed (Participants) | 68 | 79
  ARB | 13.73 (8.93) | 12.02 (8.63)
  Aldosterone Antagonists: number analyzed (Participants) | 161 | 160
  Aldosterone Antagonists | 24.16 (11.19) | 29.42 (32.68)
  Beta Blockers: number analyzed (Participants) | 285 | 284
  Beta Blockers | 30.01 (24.94) | 28.53 (25.13)
  Vasodilators (Nitrate): number analyzed (Participants) | 22 | 33
  Vasodilators (Nitrate) | 55.48 (41.64) | 48.59 (34.90)
  Vasodilators (Hydralazine): number analyzed (Participants) | 56 | 63
  Vasodilators (Hydralazine) | 133.82 (104.93) | 109.01 (87.22)
  ARNI: number analyzed (Participants) | 22 | 23
  ARNI | 10.13 (8.15) | 7.68 (4.71)

316. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 12 months
Population: as for outcome 313
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE Inhibitors: number analyzed (Participants) | 143 | 122
  ACE Inhibitors | 12.73 (13.56) | 12.41 (12.82)
  ARBs: number analyzed (Participants) | 73 | 81
  ARBs | 13.76 (9.21) | 11.90 (8.45)
  Aldosterone Antagonists: number analyzed (Participants) | 169 | 162
  Aldosterone Antagonists | 24.33 (12.17) | 29.45 (32.58)
  Beta Blockers: number analyzed (Participants) | 287 | 287
  Beta Blockers | 30.10 (24.99) | 28.19 (24.65)
  Vasodilators (Nitrate): number analyzed (Participants) | 23 | 34
  Vasodilators (Nitrate) | 56.85 (41.50) | 48.56 (34.95)
  Vasodilators (Hydralazine): number analyzed (Participants) | 60 | 68
  Vasodilators (Hydralazine) | 136.51 (99.05) | 108.74 (87.89)
  ARN Inhibitors: number analyzed (Participants) | 31 | 30
  ARN Inhibitors | 10.36 (7.57) | 7.99 (4.51)

317. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 24 months
Population: as for outcome 313
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACe Inhibitors: number analyzed (Participants) | 148 | 124
  ACe Inhibitors | 12.35 (13.36) | 12.32 (12.91)
  ARBs: number analyzed (Participants) | 78 | 83
  ARBs | 13.86 (9.10) | 11.67 (8.09)
  Aldosterone Antagonists: number analyzed (Participants) | 173 | 165
  Aldosterone Antagonists | 24.36 (12.30) | 28.98 (32.00)
  Beta Blockers: number analyzed (Participants) | 288 | 290
  Beta Blockers | 30.50 (25.15) | 27.66 (23.70)
  Vasodilators (Nitrate): number analyzed (Participants) | 24 | 39
  Vasodilators (Nitrate) | 54.81 (41.50) | 45.53 (33.30)
  Vasodilators (Hydralazine): number analyzed (Participants) | 60 | 76
  Vasodilators (Hydralazine) | 135.20 (97.01) | 102.29 (85.28)
  ARN Inhibitors: number analyzed (Participants) | 40 | 35
  ARN Inhibitors | 10.41 (7.34) | 8.52 (5.40)

318. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 3 years
Population: All available data has been reported and includes subjects on the drugs mentioned below. Not all subjects were on all thedrugs.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE Inhibitors: number analyzed (Participants) | 150 | 124
  ACE Inhibitors | 12.23 (13.29) | 12.28 (12.87)
  ARBs: number analyzed (Participants) | 81 | 87
  ARBs | 13.42 (8.88) | 11.13 (7.87)
  Aldosterone Antagonists: number analyzed (Participants) | 179 | 170
  Aldosterone Antagonists | 24.24 (11.91) | 28.97 (31.50)
  Beta Blockers: number analyzed (Participants) | 289 | 291
  Beta Blockers | 30.70 (24.66) | 27.83 (23.79)
  Vasodilators (Nitrate): number analyzed (Participants) | 27 | 43
  Vasodilators (Nitrate) | 53.37 (41.58) | 44.53 (32.50)
  Vasodilators (Hydralazine): number analyzed (Participants) | 62 | 82
  Vasodilators (Hydralazine) | 132.54 (93.88) | 101.92 (86.30)
  ARN Inhibitors: number analyzed (Participants) | 62 | 39
  ARN Inhibitors | 11.03 (7.25) | 9.68 (5.89)

319. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 4 years
Population: All available data has been reported
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE Inhibitors: number analyzed (Participants) | 152 | 124
  ACE Inhibitors | 12.10 (13.08) | 12.37 (12.89)
  ARBs: number analyzed (Participants) | 83 | 88
  ARBs | 13.28 (8.85) | 11.03 (7.83)
  Aldosterone Antagonist: number analyzed (Participants) | 183 | 171
  Aldosterone Antagonist | 24.37 (11.84) | 29.06 (31.39)
  Beta Blockers: number analyzed (Participants) | 289 | 291
  Beta Blockers | 30.59 (24.26) | 27.78 (23.80)
  Vasodilators (Nitrate): number analyzed (Participants) | 29 | 43
  Vasodilators (Nitrate) | 51.63 (40.59) | 44.59 (32.55)
  Vasodilators: number analyzed (Participants) | 64 | 83
  Vasodilators | 129.51 (93.77) | 100.74 (85.36)
  ARN Inhibitors: number analyzed (Participants) | 71 | 44
  ARN Inhibitors | 11.04 (7.29) | 9.54 (5.77)

320. Other Pre Specified Outcome: Average Dosages of GDMT
Time Frame: 5 years
Population: All available data has been reported
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
mg
  ACE Inhibitors: number analyzed (Participants) | 153 | 125
  ACE Inhibitors | 12.02 (13.03) | 12.35 (12.88)
  ARBs: number analyzed (Participants) | 84 | 88
  ARBs | 13.29 (8.78) | 11.02 (7.82)
  Aldosterone Antagonist: number analyzed (Participants) | 185 | 172
  Aldosterone Antagonist | 24.30 (11.84) | 28.99 (31.13)
  Beta Blockers: number analyzed (Participants) | 289 | 291
  Beta Blockers | 30.60 (24.16) | 27.78 (23.80)
  Vasodilators Nitrate: number analyzed (Participants) | 31 | 44
  Vasodilators Nitrate | 52.41 (40.35) | 44.28 (32.27)
  Vasodilators: number analyzed (Participants) | 65 | 84
  Vasodilators | 130.83 (93.29) | 100.07 (84.45)
  ARN Inhibitors: number analyzed (Participants) | 74 | 45
  ARN Inhibitors | 11.53 (7.34) | 9.41 (5.81)

321. Other Pre Specified Outcome: The Number of Subjects With Changes in GDMT Dosage From Baseline
Time Frame: Between baseline and 30 days
Population: Not all subjects were on all the drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors: number analyzed (Participants) | 281 | 283
  ACE-Inhibitors | 44 | 23
  Angiotensin-Receptor Blocker (ARBs): number analyzed (Participants) | 282 | 282
  Angiotensin-Receptor Blocker (ARBs) | 20 | 20
  Aldosterone Antagonists: number analyzed (Participants) | 281 | 282
  Aldosterone Antagonists | 29 | 25
  Beta Blocker: number analyzed (Participants) | 281 | 283
  Beta Blocker | 60 | 48
  Vasodilators (Nitrate): number analyzed (Participants) | 281 | 280
  Vasodilators (Nitrate) | 10 | 12
  Vasodilators (Hydralazine): number analyzed (Participants) | 281 | 282
  Vasodilators (Hydralazine) | 11 | 13

322. Other Pre Specified Outcome: The Number of Subjects With Changes in GDMT Dosage From Baseline to 6 Months
Time Frame: Between baseline and 6 months
Population: Not all subjects were on all the drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors: number analyzed (Participants) | 254 | 245
  ACE-Inhibitors | 53 | 41
  Angiotensin-Receptor Blockers (ARBs): number analyzed (Participants) | 252 | 244
  Angiotensin-Receptor Blockers (ARBs) | 35 | 27
  Aldosterone Antagonists: number analyzed (Participants) | 253 | 245
  Aldosterone Antagonists | 44 | 35
  Beta Blocker: number analyzed (Participants) | 254 | 245
  Beta Blocker | 74 | 60
  Vasodilators (Nitrate): number analyzed (Participants) | 252 | 245
  Vasodilators (Nitrate) | 14 | 18
  Vasodilators (Hydralazine): number analyzed (Participants) | 251 | 245
  Vasodilators (Hydralazine) | 15 | 20

323. Other Pre Specified Outcome: The Number of Subjects With Changes in GDMT Dosage From Baseline and 12 Months
Time Frame: Between baseline and 12 months
Population: Not all subjects were on all the drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors: number analyzed (Participants) | 219 | 203
  ACE-Inhibitors | 61 | 37
  Angiotension-Receptor Blockers (ARBs): number analyzed (Participants) | 217 | 203
  Angiotension-Receptor Blockers (ARBs) | 14 | 38
  Aldosterone Antagonists: number analyzed (Participants) | 220 | 202
  Aldosterone Antagonists | 44 | 44
  Beta Blocker: number analyzed (Participants) | 221 | 203
  Beta Blocker | 76 | 66
  Vasodilators (Nitrate): number analyzed (Participants) | 220 | 203
  Vasodilators (Nitrate) | 14 | 19
  Vasodilators (Hydralazine): number analyzed (Participants) | 220 | 203
  Vasodilators (Hydralazine) | 14 | 14

324. Other Pre Specified Outcome: The Number of Subjects With Changes in GDMT Dosage From Baseline and 24 Months
Time Frame: Between baseline and 24 months
Population: Not all subjects were on all the drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors: number analyzed (Participants) | 131 | 92
  ACE-Inhibitors | 36 | 24
  Angiotensin-Receptor Blockers (ARBs): number analyzed (Participants) | 131 | 92
  Angiotensin-Receptor Blockers (ARBs) | 29 | 21
  Aldosterone Antagonists: number analyzed (Participants) | 130 | 92
  Aldosterone Antagonists | 28 | 21
  Beta Blockers: number analyzed (Participants) | 131 | 92
  Beta Blockers | 43 | 34
  Vasodilators (Nitrate): number analyzed (Participants) | 131 | 91
  Vasodilators (Nitrate) | 7 | 11
  Vasodilators (Hydralazine): number analyzed (Participants) | 131 | 92
  Vasodilators (Hydralazine) | 10 | 14

325. Other Pre Specified Outcome: The Number and Reasons for Any Changes in GDMT and GDMT Dosage From Baseline
Time Frame: Between baseline and 3 years
Population: Not all subjects were on all the drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors: number analyzed (Participants) | 149 | 106
  ACE-Inhibitors | 44 | 25
  Angiotensin-ReceptorBlockers (ARBs): number analyzed (Participants) | 147 | 105
  Angiotensin-ReceptorBlockers (ARBs) | 40 | 26
  AldosteroneAntagonists: number analyzed (Participants) | 148 | 107
  AldosteroneAntagonists | 33 | 32
  Beta Blockers: number analyzed (Participants) | 149 | 107
  Beta Blockers | 52 | 44
  Vasodilators (Nitrate): number analyzed (Participants) | 148 | 105
  Vasodilators (Nitrate) | 20 | 9
  Vasodilators(Hydralazine): number analyzed (Participants) | 148 | 106
  Vasodilators(Hydralazine) | 17 | 12

326. Other Pre Specified Outcome: The Number and Reasons for Any Changes in GDMT and GDMT Dosage From Baseline
Time Frame: Between baseline and 4 years
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE Inhibitors: number analyzed (Participants) | 123 | 84
  ACE Inhibitors | 31 | 21
  ARBS: number analyzed (Participants) | 122 | 84
  ARBS | 39 | 27
  Aldosterone Antagonist: number analyzed (Participants) | 122 | 84
  Aldosterone Antagonist | 29 | 31
  Beta Blocker: number analyzed (Participants) | 124 | 85
  Beta Blocker | 50 | 35
  Vasodilators Nitrate: number analyzed (Participants) | 124 | 83
  Vasodilators Nitrate | 13 | 12
  Vasodilators: number analyzed (Participants) | 124 | 82
  Vasodilators | 10 | 12

327. Other Pre Specified Outcome: The Number and Reasons for Any Changes in GDMT and GDMT Dosage From Baseline
Time Frame: Between baseline and 5 years
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE Inhibitors: number analyzed (Participants) | 95 | 66
  ACE Inhibitors | 25 | 18
  ARBs: number analyzed (Participants) | 94 | 66
  ARBs | 28 | 23
  Aldosterone Antagonist: number analyzed (Participants) | 94 | 66
  Aldosterone Antagonist | 27 | 15
  Beta Blocker: number analyzed (Participants) | 95 | 66
  Beta Blocker | 40 | 33
  Vasodilators Nitrate: number analyzed (Participants) | 91 | 66
  Vasodilators Nitrate | 9 | 8
  Vasodilators: number analyzed (Participants) | 91 | 66
  Vasodilators | 6 | 13

328. Other Pre Specified Outcome: The Number of Subjects With Change in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors (Decrease > 50% or Stop) | 0 | 0
  ACE-Inhibitors (Increase > 100% or New Class) | 1 | 1
  ARB (Decrease > 50% or Stop) | 1 | 0
  ARB (Increase > 100% or New Class) | 0 | 1
  Aldosterone Antagonists (Decrease > 50% or stop) | 0 | 0
  Aldosterone Antagonists (Increase>100%orNewClass) | 2 | 2
  Beta Blockers (Decrease > 50% or Stop) | 2 | 0
  Beta Blockers (Increase >100% or New Class) | 2 | 2
  Vasodilators (Nitrate) Decrease>50% or Stop | 0 | 0
  Vasodilators (Nitrate) Increase > 100% or NewClass | 1 | 0
  Vasodilators (Hydralazine) Decrease>50% or Stop | 0 | 0
  Vasodilators(Hydralazine)Increase >100% orNewClass | 1 | 1
  ARN Inhibitors - Decrease>50% or Stop | 0 | 0
  ARN Inhibitors - Increase > 100% or NewClass | 0 | 0

329. Other Pre Specified Outcome: The Number of Subjects With Any Changes in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-I (Decrease > 50% or Stop) | 8 | 4
  ACE-I (Increase > 100% or New Class) | 6 | 4
  ARB (Decrease > 50% or Stop) | 2 | 1
  ARB (Increase > 100% or New Class) | 7 | 9
  Aldosterone Antagonists (Decrease > 50% or Stop) | 1 | 1
  Aldosterone Antagonists (Increase > 100% or NewCl) | 11 | 7
  Beta Blockers (Decrease > 50% or Stop) | 14 | 10
  Beta Blockers (Increase > 100% or New Class) | 19 | 9
  Vasodilators (Nitrate) Decrease > 50% or Stop | 0 | 0
  Vasodilators (Nitrate) Increase > 100% or NewClass | 1 | 5
  Vasodilators (Hydralazine) Decrease > 50% or Stop | 1 | 0
  Vasodilators(Hydralazine)Increase>100% orNewClass | 7 | 6
  ARN Inhibitors Decrease > 50% or Stop | 0 | 0
  ARN Inhibitors Increase > 100% or New Class | 6 | 12

330. Other Pre Specified Outcome: The Number of Subjects With Any Changes in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors Decrease > 50% or Stop | 13 | 5
  ACE-Inhibitors Increase > 100% or New Class | 9 | 8
  ARBs Decrease >50% or Stop | 3 | 2
  ARBs Increase > 100% or New Class | 13 | 12
  Aldosterone Antagonists Decrease > 50% or Stop | 2 | 2
  Aldosterone Antagonists Increase>100% or New Class | 16 | 8
  Beta Blockers Decrease > 50% or Stop | 16 | 16
  Beta Blockers Increase > 100% or New Class | 26 | 12
  Vasodilators(Nitrate) Decrease > 50% or Stop | 0 | 0
  Vasodilators(Nitrate) Increase > 100% or New Class | 3 | 6
  Vasodilators(Hydralazine) Decrease > 50% or Stop | 3 | 0
  Vasodilators(Hydralazine) Increase>100%orNewClass | 13 | 12
  ARN Inhibitors Decrease > 50% or Stop | 0 | 0
  ARN inhibitors Increase > 100% or New Class | 13 | 20

331. Other Pre Specified Outcome: The Number of Subjects With Any Changes in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors Decrease > 50% or Stop | 17 | 6
  ACE Inhibitors Increase > 100% or New Class | 14 | 11
  ARBs Decrease > 50% or Stop | 3 | 2
  ARBs Increase > 100% or New Class | 19 | 16
  Aldosterone Antagonists Decrease > 50% or Stop | 2 | 3
  Aldosterone Antagonists Increase>100% or New Class | 21 | 10
  Beta Blockers Decrease > 50% or Stop | 20 | 26
  Beta Blockers Increase > 100% or New Class | 29 | 19
  Vasodilators(Nitrate) Decrease > 50% or Stop | 0 | 1
  Vasodilators(Nitrate) Increase > 100% or New Class | 5 | 11
  Vasodilators(Hydralazine)Decrease > 50% or Stop | 6 | 1
  Vasodilators(Hydralazine) Increase>100%orNew Class | 14 | 20
  ARN Inhibitors Decrease > 50% or Stop | 0 | 0
  ARN Inhibitors Increase > 100% or New Class | 26 | 24

332. Other Pre Specified Outcome: The Number and Reasons for Any Changes in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors Decrease > 50% orStop | 19 | 7
  ACE Inhibitors Increase > 100% orNew Class | 15 | 12
  ARBs Decrease > 50% or Stop | 4 | 3
  ARBs Increase > 100% or NewClass | 22 | 19
  Aldosterone Antagonists Decrease> 50% or Stop | 3 | 5
  Aldosterone AntagonistsIncrease>100% or New Class | 27 | 14
  Beta Blockers Decrease > 50% orStop | 25 | 29
  Beta Blockers Increase > 100% orNew Class | 32 | 26
  Vasodilators(Nitrate) Decrease >50% or Stop | 0 | 1
  Vasodilators(Nitrate) Increase >100% or New Class | 6 | 13
  Vasodilators(Hydralazine)Decrease> 50% or Stop | 7 | 1
  Vasodilators(Hydralazine)Increase>100%orNew Class | 19 | 24
  ARN Inhibitors Decrease > 50% orStop | 0 | 0
  ARN Inhibitors Increase > 100% orNew Class | 45 | 29

333. Other Pre Specified Outcome: The Number and Reasons for Any Changes in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 4 years
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors Decrease > 50% orStop | 20 | 7
  ACE Inhibitors Increase > 100% orNew Class | 18 | 12
  ARBs Decrease > 50% or Stop | 5 | 3
  ARBs Increase > 100% or NewClass | 25 | 21
  Aldosterone Antagonists Decrease> 50% or Stop | 3 | 5
  Aldosterone AntagonistsIncrease>100% or New Class | 32 | 15
  Beta Blockers Decrease > 50% orStop | 29 | 32
  Beta Blockers Increase > 100% orNew Class | 35 | 26
  Vasodilators(Nitrate) Decrease >50% or Stop | 0 | 1
  Vasodilators(Nitrate) Increase >100% or New Class | 7 | 14
  Vasodilators(Hydralazine)Decrease> 50% or Stop | 7 | 3
  Vasodilators(Hydralazine)Increase>100%orNew Class | 21 | 26
  ARN Inhibitors Decrease > 50% orStop | 0 | 0
  ARN Inhibitors Increase > 100% orNew Class | 57 | 33

334. Other Pre Specified Outcome: The Number and Reasons for Any Changes in GDMT From Baseline That Result in a Greater Than 100% Increase or Greater Than 50% Decrease in Dose
Time Frame: Between baseline and 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group | Control Group
Number analyzed (Participants) | 302 | 312
Participants
  ACE-Inhibitors Decrease > 50% orStop | 20 | 7
  ACE Inhibitors Increase > 100% orNew Class | 18 | 14
  ARBs Decrease > 50% or Stop | 5 | 3
  ARBs Increase > 100% or NewClass | 26 | 22
  Aldosterone Antagonists Decrease> 50% or Stop | 4 | 5
  Aldosterone AntagonistsIncrease>100% or New Class | 33 | 16
  Beta Blockers Decrease > 50% orStop | 30 | 34
  Beta Blockers Increase > 100% orNew Class | 35 | 27
  Vasodilators(Nitrate) Decrease >50% or Stop | 0 | 1
  Vasodilators(Nitrate) Increase >100% or New Class | 9 | 15
  Vasodilators(Hydralazine)Decrease> 50% or Stop | 8 | 3
  Vasodilators(Hydralazine)Increase>100%orNew Class | 22 | 27
  ARN Inhibitors Decrease > 50% orStop | 1 | 0
  ARN Inhibitors Increase > 100% orNew Class | 62 | 34

335. Other Pre Specified Outcome: Cardiopulmonary Exercise (CPX) Testing
Description: A substudy endpoint will utilize peak oxygen consumption oxygen uptake (VO2) as a parameter for cardiopulmonary exercise testing on a total of at least 50 and up to 100 subjects.
  The CPX analysis variables are:
  * Peak VO2 (ml/kg/min) - CPX Sub-study endpoint, descriptive analysis only, not powered for statistical significance
  * Exercise duration (min)
  * Peak workload (watts)
  * Maximum heart rate during exercise (beats/min)
  * Peak VE (l/min)
  * Respiratory Exchange Ratio (RER, VCO2/VO2)
  * VE/VCO2 slope
  * Ventilatory Threshold (ml/kg/min)
  * Borg scale
  * Exercise termination reason
  * Type of exercise (treadmill vs cycling)
Time Frame: Baseline
Population: A total of 14 subjects were enrolled in the CPA sub study. However CPX data was available for only 2 subjects in the device group and 1 subject in the control group.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 2 | 1
ml/kg/min | 12.85 (0.78) | 6.00 (NA) — Data is available for only one subject. Hence Standard deviation is not applicable.

336. Other Pre Specified Outcome: Cardiopulmonary Exercise (CPX) Testing
Description: as for outcome 335
Time Frame: 12 months
Population: A total of 14 subjects participated in the CPX sub-study. CPX test data was available in 2 subjects in the device group and 1 subject in the control group.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 2 | 1
ml/kg/min | 14.50 (6.36) | 6.80 (NA) — Data available for only 1 subject. Hence Standard deviation is not possible.

337. Other Pre Specified Outcome: Cardiopulmonary Exercise (CPX) Testing: Mean Changes in Peak VO2
Description: Mean changes in peak VO2 (ml/kg/min) will be summarized at 12 months from baseline for the subset of patients who complete a CPX test at baseline and 12 months. A comparison of change from baseline between Device and Control groups will be presented.
  The CPX analysis variables are:
  * Peak VO2 (ml/kg/min) - CPX Sub-study endpoint, descriptive analysis only, not powered for statistical significance
  * Exercise duration (min)
  * Peak workload (watts)
  * Maximum heart rate during exercise (beats/min)
  * Peak VE (l/min)
  * Respiratory Exchange Ratio (RER, VCO2/VO2)
  * VE/VCO2 slope
  * Ventilatory Threshold (ml/kg/min)
  * Borg scale
  * Exercise termination reason
  * Type of exercise (treadmill vs cycling)
Time Frame: Between baseline and 12 months
Population: as for outcome 336
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | MitraClip System | Control Group
Number analyzed (Participants) | 2 | 1
ml/kg/min | 1.65 (5.59) | 0.80 (NA) — Data is available for only 1 subject.

338. Other Pre Specified Outcome: Health Economic Data
Time Frame: Through 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: COAPT IDE - 60 Months and COAPT CAS - 12 months
Description: TVT Registry Mitral module does not collect the serious adverse events for COAPT CAS group. Only AE table is being populated for the COAPT CAS group
Groups:
- COAPT CAS Group: subjects enrolled as part of the Continued Access Study with Percutaneous mitral valve repair using MitraClip System
Arm/Group | MitraClip System | Control Group | COAPT CAS Group
All-Cause Mortality (participants affected / at risk) | 167/302 | 192/312 | 46/162
Serious Adverse Events (participants affected / at risk) | 281/302 | 291/312 | 0/0
Other Adverse Events (participants affected / at risk) | 239/302 | 234/312 | 86/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip System (N=302) | Control Group (N=312) | COAPT CAS Group (N=0)
Anaemia (Blood and lymphatic system disorders) | 25 (30) | 12 (14) | 0 (0)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Anaemia of Chronic Disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 7 (8) | 2 (2) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 16 (19) | 9 (10) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 14 (16) | 21 (25) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 5 (8) | 4 (4) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 4 (4) | 5 (5) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 28 (37) | 26 (33) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 7 (9) | 7 (7) | 0 (0)
ATRIAL SEPTAL DEFECT ACQUIRED (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
ATRIAL TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 16 (17) | 28 (28) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 42 (55) | 98 (133) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 35 (45) | 39 (51) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 41 (56) | 56 (69) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 89 (136) | 105 (193) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 8 (8) | 7 (7) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 12 (14) | 20 (20) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 4 (5) | 2 (2) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
CARDIORENAL SYNDROME (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
CARDIOVASCULAR DECONDITIONING (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 6 (6) | 6 (6) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
INTRACARDIAC THROMBUS (Cardiac disorders) | 2 (2) | 3 (3) | NA
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 8 (8) | 9 (9) | NA
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 1 (1) | NA
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 3 (3) | 0 (0) | NA
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 8 (8) | 14 (15) | NA
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 (1) | 1 (1) | NA
MYOCARDIAL INFARCTION (Cardiac disorders) | 6 (6) | 6 (6) | NA
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 (3) | 0 (0) | NA
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1) | NA
PERICARDIAL EFFUSION (Cardiac disorders) | 8 (9) | 3 (3) | NA
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 (1) | 1 (1) | NA
SICK SINUS SYNDROME (Cardiac disorders) | 2 (2) | 1 (1) | NA
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 4 (4) | 0 (0) | NA
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 1 (1) | NA
TACHYARRHYTHMIA (Cardiac disorders) | 2 (2) | 0 (0) | NA
TACHYCARDIA (Cardiac disorders) | 3 (3) | 3 (3) | NA
TORSADE DE POINTES (Cardiac disorders) | 1 (1) | 1 (1) | NA
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 5 (7) | 2 (2) | NA
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 2 (2) | NA
VENTRICULAR DYSSYNCHRONY (Cardiac disorders) | 0 (0) | 2 (2) | NA
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1) | NA
VENTRICULAR FIBRILLATION (Cardiac disorders) | 5 (7) | 8 (9) | NA
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 21 (34) | 26 (40) | NA
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 0 (0) | NA
CATARACT (Eye disorders) | 2 (2) | 0 (0) | NA
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 0 (0) | NA
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1) | NA
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | NA
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (5) | 5 (5) | NA
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | NA
ACQUIRED OESOPHAGEAL WEB (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
ASCITES (Gastrointestinal disorders) | 5 (6) | 3 (5) | NA
COLITIS (Gastrointestinal disorders) | 3 (3) | 1 (1) | NA
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (2) | NA
COLONIC PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0) | NA
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 4 (4) | NA
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
DYSPHAGIA (Gastrointestinal disorders) | 7 (7) | 3 (3) | NA
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
GASTROINTESTINAL ANGIODYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 18 (21) | 20 (24) | NA
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 2 (2) | NA
INGUINAL HERNIA (Gastrointestinal disorders) | 4 (4) | 6 (6) | NA
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 2 (2) | NA
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
JEJUNITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 3 (3) | NA
MEGACOLON (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
MELAENA (Gastrointestinal disorders) | 0 (0) | 2 (2) | NA
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1) | 2 (2) | NA
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 3 (3) | NA
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
PROCTITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 6 (6) | 1 (1) | NA
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA
RECTAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
RECTAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 4 (4) | NA
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 3 (3) | NA
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (6) | 1 (1) | NA
VOLVULUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
VOMITING (Gastrointestinal disorders) | 1 (1) | 5 (7) | NA
ADVERSE DRUG REACTION (General disorders) | 2 (2) | 2 (2) | NA
ASTHENIA (General disorders) | 5 (5) | 4 (7) | NA
CATHETER SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | NA
CATHETER SITE HAEMORRHAGE (General disorders) | 4 (4) | 0 (0) | NA
CHEST DISCOMFORT (General disorders) | 1 (1) | 2 (2) | NA
CHEST PAIN (General disorders) | 10 (14) | 10 (14) | NA
DEATH (General disorders) | 12 (12) | 12 (12) | NA
DEVICE BATTERY ISSUE (General disorders) | 1 (1) | 1 (1) | NA
DEVICE DISLOCATION (General disorders) | 7 (7) | 0 (0) | NA
DEVICE ELECTRICAL FINDING (General disorders) | 4 (4) | 2 (3) | NA
DEVICE LEAD DAMAGE (General disorders) | 1 (1) | 0 (0) | NA
DEVICE LEAD ISSUE (General disorders) | 1 (1) | 0 (0) | NA
DEVICE MALFUNCTION (General disorders) | 6 (6) | 0 (0) | NA
DRUG INTOLERANCE (General disorders) | 0 (0) | 1 (1) | NA
EXERCISE TOLERANCE DECREASED (General disorders) | 0 (0) | 1 (1) | NA
FATIGUE (General disorders) | 1 (1) | 2 (2) | NA
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (2) | 0 (0) | NA
HERNIA (General disorders) | 2 (2) | 0 (0) | NA
HERNIA OBSTRUCTIVE (General disorders) | 1 (1) | 0 (0) | NA
MEDICAL DEVICE COMPLICATION (General disorders) | 2 (2) | 2 (2) | NA
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 3 (3) | NA
NON-CARDIAC CHEST PAIN (General disorders) | 7 (8) | 7 (10) | NA
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 4 (4) | NA
PYREXIA (General disorders) | 5 (6) | 2 (3) | NA
SUDDEN CARDIAC DEATH (General disorders) | 2 (2) | 1 (1) | NA
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0) | NA
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3) | 1 (1) | NA
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 4 (4) | 3 (3) | NA
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 1 (1) | NA
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | NA
HEPATIC MASS (Hepatobiliary disorders) | 0 (0) | 1 (1) | NA
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | NA
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | NA
HEART TRANSPLANT REJECTION (Immune system disorders) | 2 (2) | 1 (1) | NA
IMMUNOSUPPRESSION (Immune system disorders) | 0 (0) | 1 (1) | NA
TRANSPLANT REJECTION (Immune system disorders) | 1 (2) | 0 (0) | NA
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | NA
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0) | NA
ACQUIRED IMMUNODEFICIENCY SYNDROME (Infections and infestations) | 0 (0) | 1 (1) | NA
BACTERAEMIA (Infections and infestations) | 5 (6) | 0 (0) | NA
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | NA
BRONCHITIS (Infections and infestations) | 2 (2) | 4 (4) | NA
BRONCHITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1) | NA
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | NA
CELLULITIS (Infections and infestations) | 10 (10) | 6 (7) | NA
CLOSTRIDIAL INFECTION (Infections and infestations) | 2 (2) | 1 (1) | NA
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (3) | 5 (7) | NA
CYSTITIS (Infections and infestations) | 2 (2) | 0 (0) | NA
DEVICE RELATED INFECTION (Infections and infestations) | 2 (2) | 3 (5) | NA
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | NA
DIVERTICULITIS (Infections and infestations) | 5 (6) | 3 (3) | NA
EMPHYSEMATOUS CYSTITIS (Infections and infestations) | 1 (1) | 1 (1) | NA
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1) | NA
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | NA
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | NA
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | NA
FUNGAEMIA (Infections and infestations) | 1 (1) | 0 (0) | NA
GANGRENE (Infections and infestations) | 2 (2) | 0 (0) | NA
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 2 (2) | NA
HERPES ZOSTER (Infections and infestations) | 3 (3) | 1 (1) | NA
IMPLANT SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | NA
INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
INFLUENZA (Infections and infestations) | 4 (4) | 6 (6) | NA
INFUSION SITE CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | NA
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | NA
LOBAR PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | NA
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | NA
OESOPHAGEAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | NA
OSTEOMYELITIS (Infections and infestations) | 2 (2) | 1 (1) | NA
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | NA
PERITONITIS (Infections and infestations) | 2 (2) | 1 (1) | NA
PNEUMONIA (Infections and infestations) | 27 (33) | 28 (32) | NA
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | NA
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 1 (1) | NA
PNEUMONIA NECROTISING (Infections and infestations) | 1 (1) | 0 (0) | NA
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 (0) | 1 (1) | NA
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | NA
POST VIRAL FATIGUE SYNDROME (Infections and infestations) | 0 (0) | 1 (1) | NA
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | NA
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 1 (1) | NA
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | NA
SEPSIS (Infections and infestations) | 18 (20) | 13 (15) | NA
SEPSIS SYNDROME (Infections and infestations) | 1 (1) | 0 (0) | NA
SEPTIC SHOCK (Infections and infestations) | 6 (6) | 9 (9) | NA
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 2 (2) | 2 (2) | NA
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 1 (1) | NA
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (2) | NA
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | NA
TRACHEOBRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | NA
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | NA
URINARY TRACT INFECTION (Infections and infestations) | 4 (7) | 5 (6) | NA
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | NA
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 1 (1) | 0 (0) | NA
UROSEPSIS (Infections and infestations) | 3 (3) | 4 (4) | NA
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | NA
ANAESTHETIC COMPLICATION PULMONARY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
CARDIAC VALVE REPLACEMENT COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | NA
COMPLICATIONS OF TRANSPLANTED HEART (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | NA
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | NA
FACE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
FALL (Injury, poisoning and procedural complications) | 14 (14) | 15 (15) | NA
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | NA
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | NA
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
GASTROENTERITIS RADIATION (Injury, poisoning and procedural complications) | 1 (7) | 0 (0) | NA
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | NA
HIP FRACTURE (Injury, poisoning and procedural complications) | 6 (6) | 8 (8) | NA
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | NA
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | NA
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | NA
POCKET EROSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | NA
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 3 (5) | NA
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | NA
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | NA
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | NA
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | NA
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
RENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | NA
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | NA
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | NA
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | NA
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | NA
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | NA
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | NA
VENA CAVA INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 3 (4) | 0 (0) | NA
CARDIAC ENZYMES INCREASED (Investigations) | 0 (0) | 1 (1) | NA
CARDIAC OUTPUT DECREASED (Investigations) | 0 (0) | 1 (1) | NA
CATHETERISATION CARDIAC (Investigations) | 1 (1) | 0 (0) | NA
COLONOSCOPY (Investigations) | 1 (1) | 0 (0) | NA
DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 1 (1) | 0 (0) | NA
EJECTION FRACTION DECREASED (Investigations) | 3 (3) | 1 (1) | NA
ELECTROCARDIOGRAM AMBULATORY ABNORMAL (Investigations) | 0 (0) | 1 (1) | NA
ELECTROCARDIOGRAM QRS COMPLEX PROLONGED (Investigations) | 0 (0) | 1 (1) | NA
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 1 (1) | NA
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 1 (1) | 0 (0) | NA
ENTEROCOCCUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | NA
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0) | NA
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0) | NA
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 0 (0) | 1 (1) | NA
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 3 (3) | NA
LABORATORY TEST ABNORMAL (Investigations) | 0 (0) | 1 (1) | NA
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 (2) | 1 (1) | NA
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 1 (1) | NA
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0) | NA
URINE OUTPUT DECREASED (Investigations) | 1 (1) | 0 (0) | NA
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | NA
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | NA
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | NA
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | NA
FLUID OVERLOAD (Metabolism and nutrition disorders) | 6 (8) | 5 (5) | NA
GOUT (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | NA
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | NA
HYPERKALAEMIA (Metabolism and nutrition disorders) | 7 (7) | 6 (7) | NA
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | NA
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 (6) | 5 (6) | NA
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | NA
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | NA
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | NA
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | NA
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | NA
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | NA
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | NA
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | NA
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | NA
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | NA
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | NA
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | NA
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
ANGIOSARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | NA
BONE SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | NA
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | NA
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
CAROTID ARTERY DISEASE (Nervous system disorders) | 2 (2) | 0 (0) | NA
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 1 (1) | NA
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | NA
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 4 (4) | 0 (0) | NA
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 16 (17) | 11 (12) | NA
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | NA
CONVULSION (Nervous system disorders) | 1 (1) | 1 (1) | NA
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 (0) | 1 (1) | NA
DIZZINESS (Nervous system disorders) | 3 (3) | 2 (2) | NA
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1) | 0 (0) | NA
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0) | NA
EMBOLIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | NA
ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 4 (4) | NA
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0) | NA
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | NA
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 2 (2) | NA
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1) | NA
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | NA
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 1 (1) | NA
INTRACRANIAL HYPOTENSION (Nervous system disorders) | 1 (1) | 0 (0) | NA
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 3 (3) | NA
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 2 (2) | NA
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 2 (2) | NA
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 1 (1) | NA
PRESYNCOPE (Nervous system disorders) | 3 (3) | 0 (0) | NA
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | NA
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 3 (3) | 2 (2) | NA
SYNCOPE (Nervous system disorders) | 14 (16) | 22 (24) | NA
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1) | NA
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 (4) | 5 (5) | NA
VERTEBRAL ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (1) | NA
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 2 (2) | NA
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0) | NA
DISORIENTATION (Psychiatric disorders) | 0 (0) | 1 (1) | NA
MENTAL STATUS CHANGES (Psychiatric disorders) | 10 (10) | 4 (5) | NA
PANIC ATTACK (Psychiatric disorders) | 1 (1) | 0 (0) | NA
AZOTAEMIA (Renal and urinary disorders) | 1 (1) | 3 (5) | NA
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
HAEMATURIA (Renal and urinary disorders) | 5 (6) | 4 (5) | NA
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2) | 1 (1) | NA
NEPHROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
RENAL FAILURE (Renal and urinary disorders) | 6 (6) | 10 (10) | NA
RENAL FAILURE ACUTE (Renal and urinary disorders) | 41 (49) | 51 (60) | NA
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 12 (15) | 20 (21) | NA
RENAL IMPAIRMENT (Renal and urinary disorders) | 3 (3) | 5 (5) | NA
RENAL MASS (Renal and urinary disorders) | 0 (0) | 2 (2) | NA
URINARY RETENTION (Renal and urinary disorders) | 5 (6) | 1 (1) | NA
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 2 (2) | NA
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | NA
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (5) | NA
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 14 (14) | NA
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | NA
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | NA
BRONCHIAL SECRETION RETENTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
CHRONIC OBSTRUCTIVE PULMONARY DISORDER (Respiratory, thoracic and mediastinal disorders) | 10 (18) | 10 (16) | NA
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 16 (18) | NA
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | NA
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1) | NA
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | NA
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | NA
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | NA
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
LARYNGEAL HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
MEDIASTINAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 14 (18) | NA
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | NA
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | NA
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | NA
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | NA
RALES (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | NA
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | NA
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 19 (19) | NA
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | NA
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
DIGITAL ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | NA
AORTIC SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0) | NA
CARDIAC PACEMAKER BATTERY REPLACEMENT (Surgical and medical procedures) | 1 (1) | 1 (1) | NA
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 1 (1) | 1 (1) | NA
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 (1) | 1 (1) | NA
GASTRECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | NA
HEART TRANSPLANT (Surgical and medical procedures) | 0 (0) | 1 (1) | NA
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1) | NA
IMPLANTABLE DEFIBRILLATOR INSERTION (Surgical and medical procedures) | 1 (1) | 0 (0) | NA
IMPLANTABLE DEFIBRILLATOR REPLACEMENT (Surgical and medical procedures) | 2 (3) | 0 (0) | NA
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1) | NA
MEDICAL DEVICE CHANGE (Surgical and medical procedures) | 1 (1) | 0 (0) | NA
PERCUTANEOUS CORONARY INTERVENTION (Surgical and medical procedures) | 1 (1) | 0 (0) | NA
SPINAL FUSION SURGERY (Surgical and medical procedures) | 2 (2) | 0 (0) | NA
ANGIOPATHY (Vascular disorders) | 0 (0) | 1 (1) | NA
AORTIC ANEURYSM (Vascular disorders) | 2 (2) | 2 (2) | NA
AORTIC STENOSIS (Vascular disorders) | 2 (2) | 2 (2) | NA
ARTERIOSCLEROSIS (Vascular disorders) | 3 (3) | 2 (2) | NA
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 3 (3) | NA
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | NA
HAEMATOMA (Vascular disorders) | 5 (5) | 1 (1) | NA
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 1 (1) | NA
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0) | NA
HYPOTENSION (Vascular disorders) | 24 (27) | 18 (19) | NA
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 1 (1) | NA
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 (0) | 1 (1) | NA
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 (3) | 2 (2) | NA
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | NA
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (2) | 3 (3) | NA
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0) | NA
PERIPHERAL ISCHAEMIA (Vascular disorders) | 4 (4) | 2 (2) | NA
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 2 (2) | 1 (1) | NA
SHOCK (Vascular disorders) | 2 (2) | 1 (1) | NA
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 1 (1) | NA
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
ACUTE RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | NA
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1) | NA
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 0 (0) | NA
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 (1) | 0 (0) | NA
CARDIAC PERFORATION (Cardiac disorders) | 1 (1) | 0 (0) | NA
CHRONIC LEFT VENTRICULAR FAILURE (Cardiac disorders) | 3 (4) | 2 (2) | NA
LOW CARDIAC OUTPUT SYNDROME (Cardiac disorders) | 1 (1) | 1 (1) | NA
MITRAL VALVE DISEASE (Cardiac disorders) | 0 (0) | 2 (2) | NA
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 2 (2) | NA
BLINDNESS UNILATERAL (Eye disorders) | 1 (1) | 0 (0) | NA
EYE HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | NA
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 1 (1) | NA
DUODENAL VASCULAR ECTASIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
GASTROINTESTINAL VASCULAR MALFORMATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
OESOPHAGITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
CYST (General disorders) | 1 (1) | 0 (0) | NA
DEVICE OCCLUSION (General disorders) | 0 (0) | 1 (1) | NA
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0) | NA
IMPLANT SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | NA
ISCHAEMIC ULCER (General disorders) | 1 (1) | 0 (0) | NA
MASS (General disorders) | 0 (0) | 1 (1) | NA
THROMBOSIS IN DEVICE (General disorders) | 2 (2) | 1 (1) | NA
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
CARDIAC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
AMERICAN TRYPANOSOMIASIS (Infections and infestations) | 0 (0) | 1 (1) | NA
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | NA
CORONA VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | NA
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | NA
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1) | 0 (0) | NA
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1) | NA
TRACHEOBRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | NA
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
BLADDER INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | NA
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
LIP INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
ANTICOAGULATION DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 1 (1) | 2 (2) | NA
BARIUM SWALLOW ABNORMAL (Investigations) | 1 (1) | 0 (0) | NA
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 1 (1) | 0 (0) | NA
CARDIAC MONITORING (Investigations) | 0 (0) | 1 (1) | NA
NOROVIRUS TEST POSITIVE (Investigations) | 1 (1) | 1 (1) | NA
RESPIRATORY SYNCYTIAL VIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0) | NA
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
FRACTURE MALUNION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | NA
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
ONCOLOGIC COMPLICATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | NA
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
DURAL FISTULA (Nervous system disorders) | 1 (1) | 0 (0) | NA
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | NA
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
RENAL DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
PROSTATIC HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | NA
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
PULMONARY HILUM MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
TRACHEOMALACIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
CUTIS LAXA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
PANNICULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
HYPERTENSION (Vascular disorders) | 2 (2) | 2 (2) | NA
THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1) | NA
VENOUS OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | NA
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1) | NA
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 0 (0) | NA
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0) | NA
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | NA
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | NA
BLADDER MASS (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
PERIPHERAL EMBOLISM (Vascular disorders) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip System (N=302) | Control Group (N=312) | COAPT CAS Group (N=162)
ANAEMIA (Blood and lymphatic system disorders) | 18 (19) | 20 (22) | 0 (0)
ANAEMIA FOLATE DEFICIENCY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 0 (0)
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
MACROCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 (10) | 6 (6) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 3 (3) | 6 (6) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 23 (28) | 16 (19) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 2 (4) | 4 (4) | 0 (0)
ATRIAL SEPTAL DEFECT ACQUIRED (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 6 (6) | 9 (10) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 5 (5) | 7 (8) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 5 (5) | 6 (7) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 16 (17) | 21 (31) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CYANOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
INTRACARDIAC THROMBUS (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 9 (11) | 4 (4) | 0 (0)
MITRAL VALVE STENOSIS (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 6 (7) | 3 (4) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 5 (5) | 2 (2) | 0 (0)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 18 (20) | 8 (8) | 0 (0)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 1 (2) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 4 (5) | 2 (2) | 0 (0)
THYROIDITIS (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
BLEPHARITIS (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 3 (6) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL VASCULAR OCCLUSION (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
ABDOMINAL MASS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (10) | 5 (8) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 3 (4) | 0 (0)
ASCITES (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 7 (7) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRIC POLYPS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 7 (8) | 8 (11) | 0 (0)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL HYPOMOTILITY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PAROTID GLAND INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
POOR DENTAL CONDITION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0)
SALIVARY GLAND DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
TONGUE ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 5 (6) | 14 (16) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 10 (10) | 10 (11) | 0 (0)
APPLICATION SITE PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 7 (10) | 7 (8) | 0 (0)
CATHETER SITE DISCHARGE (General disorders) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 3 (3) | 0 (0) | 0 (0)
CATHETER SITE HAEMORRHAGE (General disorders) | 16 (16) | 3 (3) | 0 (0)
CATHETER SITE INFLAMMATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE PAIN (General disorders) | 2 (2) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 4 (5) | 3 (3) | 0 (0)
CHEST PAIN (General disorders) | 8 (13) | 13 (15) | 0 (0)
CYST (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE BATTERY ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE CAPTURING ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE ELECTRICAL FINDING (General disorders) | 1 (1) | 2 (2) | 0 (0)
DEVICE INFUSION ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE LEAD DAMAGE (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE MALFUNCTION (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE STIMULATION ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
EXERCISE TOLERANCE DECREASED (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 14 (18) | 9 (9) | 0 (0)
GENERALISED OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTHERMIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
INFUSION SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 0 (0) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0)
MEDICAL DEVICE COMPLICATION (General disorders) | 0 (0) | 2 (2) | 0 (0)
MUCOSAL HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 7 (10) | 8 (12) | 0 (0)
OEDEMA (General disorders) | 4 (4) | 3 (3) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 15 (16) | 13 (18) | 0 (0)
PELVIC MASS (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 4 (4) | 2 (2) | 0 (0)
ULCER (General disorders) | 1 (1) | 0 (0) | 0 (0)
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
VESSEL PUNCTURE SITE HAEMORRHAGE (General disorders) | 2 (2) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
HEPATIC CONGESTION (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 8 (10) | 7 (8) | 0 (0)
CANDIDIASIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 5 (7) | 5 (5) | 0 (0)
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
CYSTITIS KLEBSIELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
EAR INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
ENDOCARDITIS ENTEROCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
INCISION SITE ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTED BITES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 7 (7) | 1 (1) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 7 (7) | 3 (3) | 0 (0)
ONYCHOMYCOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
OTITIS MEDIA ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 16 (18) | 13 (14) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (14) | 9 (10) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 23 (32) | 19 (19) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
VIRAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
AGITATION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
EAR ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
EAR INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ENDOTRACHEAL INTUBATION COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
FACE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 20 (21) | 21 (26) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FROSTBITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 12 (15) | 9 (9) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
OPEN WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL DIARRHOEA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
POST PROCEDURAL HYPOTHYROIDISM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKIN WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
URETHRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
AMYLASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
ANTIBIOTIC RESISTANT STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 2 (3) | 0 (0) | 0 (0)
ANTICOAGULATION DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 2 (3) | 0 (0) | 0 (0)
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 2 (2) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 6 (7) | 3 (3) | 0 (0)
BLOOD CREATINE MB PHOSPHOKINASE INCREASED (Investigations) | 8 (8) | 9 (12) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 9 (10) | 6 (7) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
BLOOD PRESSURE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 2 (2) | 3 (3) | 0 (0)
CARCINOEMBRYONIC ANTIGEN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ENZYMES INCREASED (Investigations) | 2 (3) | 1 (1) | 0 (0)
CARDIAC INDEX DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
CARDIAC OUTPUT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
COMPUTERISED TOMOGRAM ABDOMEN ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 1 (1) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 3 (3) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM CHANGE (Investigations) | 0 (0) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 2 (2) | 3 (3) | 0 (0)
FIBRIN D DIMER INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HAEMATOLOGY TEST ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEART RATE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
HELICOBACTER TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 2 (2) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 4 (4) | 4 (4) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 4 (5) | 0 (0)
N-TERMINAL PROHORMONE BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
OCCULT BLOOD POSITIVE (Investigations) | 1 (1) | 0 (0) | 0 (0)
OXYGEN CONSUMPTION DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 3 (3) | 0 (0)
PROTHROMBIN TIME PROLONGED (Investigations) | 0 (0) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
TROPONIN I INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 5 (5) | 11 (11) | 0 (0)
ULTRASOUND ABDOMEN NORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 2 (2) | 6 (7) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 1 (2) | 0 (0)
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 8 (10) | 0 (0)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 8 (10) | 5 (5) | 0 (0)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 11 (14) | 12 (16) | 0 (0)
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 17 (18) | 10 (10) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10 (13) | 12 (13) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (7) | 14 (16) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
LACTOSE INTOLERANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NECK MASS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (10) | 0 (0)
RENAL OSTEODYSTROPHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PARAPROTEINAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0)
DEMENTIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 18 (24) | 15 (18) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 6 (6) | 3 (3) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
ESSENTIAL TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (4) | 5 (5) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 4 (5) | 2 (2) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
MYOCLONUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARKINSONISM (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PHANTOM PAIN (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 3 (3) | 7 (8) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 8 (8) | 10 (13) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
VASCULAR DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 4 (4) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
DELIRIUM (Psychiatric disorders) | 3 (3) | 4 (5) | 0 (0)
DEPRESSION (Psychiatric disorders) | 4 (4) | 4 (4) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 6 (6) | 3 (3) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 8 (8) | 3 (3) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
BLADDER SPASM (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 5 (5) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 13 (13) | 7 (7) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
PYURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
RENAL CYST (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 8 (8) | 7 (7) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 27 (30) | 29 (40) | 0 (0)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 9 (9) | 4 (4) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 3 (3) | 4 (5) | 0 (0)
RENAL INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL MASS (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 8 (8) | 4 (4) | 0 (0)
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
BREAST INFLAMMATION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
BREAST MASS (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
GYNAECOMASTIA (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (14) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 27 (39) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
DYSPNOEA PAROXYSMAL NOCTURNAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 11 (11) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 13 (13) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CUTIS LAXA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC PACEMAKER BATTERY REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
MEDICAL DEVICE BATTERY REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
RENAL STONE REMOVAL (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ROUTINE HEALTH MAINTENANCE (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (4) | 6 (7) | 0 (0)
HYPOTENSION (Vascular disorders) | 35 (38) | 29 (33) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
ORTHOSTATIC HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
SUBCLAVIAN ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
CHRONIC LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
DEAFNESS BILATERAL (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
EUTHYROID SICK SYNDROME (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
CHALAZION (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
EPISCLERITIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
MYOPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHANGE OF BOWEL HABIT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 13 (14) | 10 (13) | 0 (0)
DIVERTICULUM OESOPHAGEAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FAECALOMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC CYST (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE OCCLUSION (General disorders) | 1 (1) | 0 (0) | 0 (0)
EARLY SATIETY (General disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE TONSILLITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
WOUND INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SKIN INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
BLOOD SODIUM ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
CARDIAC PACEMAKER EVALUATION (Investigations) | 1 (1) | 0 (0) | 0 (0)
POSITRON EMISSION TOMOGRAM ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
SERUM FERRITIN DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
SIMPLEX VIRUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2) | 0 (0)
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERSOMNIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
GENITAL LESION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESTRICTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
EXTREMITY NECROSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
LABILE HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ASD Closure Following Transseptal Catheterization (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (3) — This falls under Additional procedures for the TVT registry Mitral module
Mitral Valve Reintervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 4 (4) — Falls under additional procedure for the TVT Registry module
Unplanned Other Cardiac Surgery or Intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 7 (8)
Other Device Related Event (General disorders) | 0 (0) | 0 (0) | 3 (3)
Single Leaflet Device Attachment (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemic Stroke (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Readmission (Cardiac disorders) | 0 (0) | 0 (0) | 18 (20)
Heart Failure Readmission (Cardiac disorders) | 0 (0) | 0 (0) | 38 (55)
Non Cardiac Readmission (Cardiac disorders) | 0 (0) | 0 (0) | 43 (76)
New Requirement for Dialysis (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Mitral Leaflet Injury (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Bleeding at Access Site (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
GU Bleed (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Life threatening Bleeding (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Major Bleeding Event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Major Vascular Complications (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Other Bleed (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT01626079/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT01626079/SAP_001.pdf